#### The GlaxoSmithKline group of companies

208749

| Division | : Worldwide Development |
|---|---|
| Information Type : Reporting and Analysis Plan (RAP) | |

Title : Reporting and Analysis Plan for A Pilot Open-Label Clinical Trial Evaluating the Safety and Efficacy of Autologous T Cells Expressing Enhanced TCRs Specific for NY-ESO-1 in Subjects with Stage IIIb or Stage IV Non-Small Cell Lung Cancer (NSCLC)

Compound Number : GSK3377794

Effective Date : Refer to Document Date

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol GSK208749
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Author | Date |
|---------------------------------------------|-------------|
| PPD | 16 CED 2020 |
| Statistician (Oncology Clinical Statistics) | 16-SEP-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

208749

# **RAP Team Reviewer (Method: Email)**

| Reviewer | Date |
|---|---|
| PPD | |
| VP Clinical Development, Cell & Gene Therapy (Oncology Clinical) | 17-SEP-2020 |
| PPD | 16-SEP-2020 |
| Programming Manager (Oncology Clinical Programming) | 10-SEF-2020 |
| PPD | |
| Clinical Biomarker Lead (Translational Research and Development) | 16-SEP-2020 |
| PPD | |
| Quantitative Clinical Pharmacology Director (Oncology CPMS) | 16-SEP-2020 |

# Clinical Statistics and Clinical Programming Line Approvals: (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| Statistics Director (Oncology Clinical Statistics) On behalf of PPD (Senior Statistics Director Oncology Clinical Statistics) | Refer to Document<br>Date |
| Programming Manager (Oncology Clinical Programming) | Refer to Document<br>Date |

208749

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 7 |
| 2. | SUM | MARY OF KEY PROTOCOL INFORMATION | 8 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 9 |
| | 2.3. | Study Design | 11 |
| | 2.4. | Statistical Analyses | |
| 3. | PI AN | INED ANALYSES | 13 |
| Ο. | 3.1. | Primary Analyses | |
| | 3.2. | Final Analyses | |
| 4. | ANAL | YSIS POPULATIONS | 13 |
| | 4.1. | Protocol Deviations | |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| Ο. | | VENTIONS | 15 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicenter Studies | 16 |
| | 5.4. | Examination of Covariates, Other Strata, and Subgroups | 16 |
| | 5.5. | Multiple Comparison and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 16 |
| | | Conventions | 10 |
| 6. | STUE | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | |
| | 6.2. | Disposition of Participants | |
| | 6.3. | Protocol Deviations | |
| | 6.4. | Demographic and Baseline Characteristics | |
| | 6.5. | Study Treatment Exposure | |
| | 6.6. | Anti-Cancer Therapy and Surgery | |
| | 6.7. | Concomitant Medications | 20 |
| <b>7</b> . | | CACY ANALYSES | |
| | 7.1. | Secondary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent Events | |
| | 7.0 | 7.1.5. Statistical Analyses / Methods | |
| | 7.2. | Exploratory Efficacy Analyses | |
| | | 7.2.1. Overall Survival | |
| | | • | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.5. Statistical Analyses / Methods | |
| 0 | CAEE | TV ANALYSES | 21 |

| | 8.1. | Adverse | Events Analyses | 31 |
|---|---|---|---|---|
| | 8.2. | | Events of Special Interest Analyses | |
| | | 8.2.1. | Cytokine Release Syndrome (CRS) and Graft versus Host | |
| | | | Disease (GvHD) | |
| | 8.3. | | and Serious Adverse Events | |
| | 8.4. | | _aboratory Analyses | |
| | | 8.4.1. | Analyses of Liver Function Tests (LFT) | |
| | 8.5. | | afety Analyses | |
| | | 8.5.1. | Performance Status | |
| | | 8.5.2. | ECG | |
| | | 8.5.3. | Vital Signs | |
| | | 8.5.4. | Pregnancies | 39 |
| | | 8.5.5. | Replication Competent Lentivirus (RCL) and Persistence of NY-ESO-1 <sup>c259</sup> T | 39 |
| 9. | BIOM | ARKER AI | NALYSES | 40 |
| | 9.1. | | ory Biomarker Analyses | |
| | | 9.1.1. | Endpoint / Variables | |
| | | 9.1.2. | Summary Measure | |
| | | • | 9.1.2.1. Persistence of NY-ESO-1 <sup>c259</sup> T | 40 |
| | | | 9.1.2.2. Cytokines | |
| | | 9.1.3. | Population of Interest | |
| 10. | PHAR | MAKOKIN | NETIC ANALYSES | 41 |
| 11. | POPU | LATION F | PHARMACOKINETIC (POPPK) ANALYSES | 41 |
| 12. | PHAR | MACOKIN | NETIC / PHARMACODYNAMIC ANALYSES | 42 |
| 13. | REFE | RENCES. | | 43 |
| 14. | APPE | | | 44 |
| | 14.1. | Appendix | x 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | 14.2. | Appendix | x 2: Schedule of Activities | 45 |
| | | 14.2.1. | Protocol Defined Schedule of Events Interventional Phase | 45 |
| | | 14.2.2. | Protocol Schedule of Events Interventional Phase II | |
| | | 14.2.2. | | 51 |
| | | 14.2.3. | Protocol Defined Schedule of Events Long Term Follow- | EG |
| | 44.0 | A no o o di | up | |
| | 14.3.<br>14.4. | | x 3: Assessment Windows | 56 |
| | 14.4. | | x 4: Study Phases and Treatment Emergent Adverse | E0 |
| | | | Other Disease | |
| | | 14.4.1. | | |
| | | | 14.4.1.1. Study Phases for Concomitant Medications | |
| | | 44.40 | 14.4.1.2. Study Phases for Anti-Cancer Therapy/Surgery | |
| | 44.5 | 14.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 14.5. | | x 5: Data Display Standards & Handling Conventions | 60 |
| | | 14.5.1. | Reporting Process | |
| | 440 | 14.5.2. | Reporting Standards | |
| | 14.6. | | x 6: Derived and Transformed Data | 62 |
| | | 1/1 16 1 | LEADARD | ₩') |

| | 14.6.2. | Study Population | |
|---|---|---|---|
| | 14.6.3. | Efficacy | 63 |
| | 14.6.4. | Safety | |
| 14.7. | Appendix | 7: Reporting Standards for Missing Data | 65 |
| | | Premature Withdrawals | |
| | | Handling of Missing Data | |
| | | 14.7.2.1. Handling of Missing and Partial Dates | |
| 14.8. | Appendix | x 8: Values of Potential Clinical Importance | |
| | | Laboratory Values | |
| | | ECG Parameters | |
| | | Vital Signs | |
| 14.9. | | c 9: Abbreviations & Trade Marks | |
| | 14.9.1. | Abbreviations | |
| | 14.9.2. | | |
| 14.10. | Appendix | c 10: List of Data Displays | |
| | | Mock Example Shell Referencing | |
| | | Data Display Numbering | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Biomarker Tables. | |
| | | .Biomarker Figures | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 14.11. | | x 11: Example Mock Shells for Data Displays | |
| | | POP_T1 Exposure Mock-Up Summary | |
| | | EFF_F1 Spider Plot Mock-Up Figure | |
| | | SAFE_F1 Prior Therapy Mock-Up Figure | |
| | | SAFE_F2 Study Duration Mock Up Figure | |
| | | BIO_F3 Persistence Profile Mock-Up Figure | |
| | | BIO_F4 Cytokine Spider Plot Mock-Up Figure | |
| | | BIO_F5 Cytokine Box Plot Figure | |
| | | SAFE_L1 CRS Mock-Up Listing | |
| | | BIO_T1 Summary of Peak Persistence | |
| | | .BIO_T2 Summary of Time to Peak Persistence | |
| | | .SAFE T3 Summary of Replication Competent Lentivirus | 122 |
| | | Positive | 123 |
| | 14 11 12 | .BIO_L1 Listing of Persistence | 124 |
| | | .POP L1 Listing of Exposure to T-cell Infusion | |
| | | .POP_L2 Listing of Exposure to Cyclophosphamide/Mesna | |
| | | .POP_L3 Listing of Leukapheresis, Lymphodepletion, and | 121 |
| | 14.11.10 | T-cell Infusion Dates | 128 |
| | 14 11 16 | .POP_L4 Listing of Disease Characteristics at Screening | |
| | | .POP_L5 Subject Status Mock-Up Listing | |
| | | .EFF_T1 Summary of Time to Response by Investigator | 101 |
| | 17.11.10 | (RECIST 1.1 Criteria) | 132 |
| | 14 11 10 | .SAFE_T1 Summary of Time to Resolution | |
| | | .POP_T2 Summary of Subject Status | |
| | | .POP_12 Summary of Subject Status | |
| | 17.11.41 | . To To Juli linary of Judicol Jlalus- Eliu of Jlauy | 100 |

# 208749 | Statistical Analysis Plan RAP 02 Oct 2020 | TMF-2069301 | 1.0


| | 208748 |
|---------------------------------------------------------|----------|
| 14.11.22.SAFE_L2 Listing of Symptoms, Concomitant Medic | cations, |
| and Procedures Related to Cytokine Release Sync | drome136 |
| 14.11.23.BIO L2 Listing of Immunohistochemistry Data | 137 |
| 14.12. Appendix 12: Combined Preferred Terms | 138 |
| 14.13. Appendix 13: AE Collapsing Rules | 140 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronol | ogy: | |
|---|---|---|
| ADP-0011-004 | 08-JUN-2015 | Original protocol was provided by Adaptimmune |
| ADP-0011-004 08-<br>Amendment 01 | 08-AUG-2016 | This amendment was performed to address questions and comments from Institutional Review Boards and Regulatory Authorities. Additionally, revisions were made based on emerging data from Adaptimmune's clinical program and due to Adaptimmune's newly developed protocol template. Appendix 8 in the protocol contains a summary of and rationale for all revisions for Amendment 01. |
| | | Key revisions included the following: |
| | | Changed phase of trial from Phase I/II to Pilot |
| | | Revised Background and Study Rationale sections to minimize information already provided in the NY-ESO-1c259T Investigator Brochure |
| | | Revised primary, secondary, and exploratory endpoints to better characterize the safety and efficacy evaluations, and correlative studies to be performed in this study |
| | | Changed lymphodepleting chemotherapy regimen from cyclophosphamide alone to cyclophosphamide and fludarabine based on emerging data from our ongoing clinical program |
| | | Removed HLA and antigen expression screening since these tests will be performed in Adaptimmune's Screening Protocol (ADP-0000-001) |
| | | Revised inclusion/exclusion criteria to provide more clarity on participant population |
| | | Added guidance on second T cell infusion, including eligibility criteria and Schedule of Procedures table |
| | | Added text around the administration of cyclophosphamide and fludarabine, including dose adjustments, prophylactic and supportive treatments |
| | | Removed irRC criteria for tumor response assessments |
| | | Added several sections on supportive care guidance, including infection, hematologic and blood product support, autoimmunity, GVHD, and pancytopenia |

208749

| GSK208749<br>Amendment 02 | 16-July-2017 | Subsequent to the licensing of Adaptimmune product NY-ESO by GSK, the purpose of this protocol amendment is to: |
|---|---|---|
| | | Delete or replace references to Adaptimmune or its staff with that of GlaxoSmithKline (GSK) and its authorized agents to align with the change of sponsorship; |
| | | Make administrative changes to align with GSK processes and procedures; |
| | | Update language relating to serious adverse event (SAE) reporting and safety monitoring. |
| | | - Changes to lymphodepletion regimen throughout |
| GSK208749<br>Amendment 03 | 17-October-<br>2018 | Changes made to the protocol were requested by the FDA as a result of safety events which included 2 reports of Guillain-Barré syndrome in participants who have received chemotherapy and GSK3377794 during clinical trials. |
| GSK208749<br>Amendment 04 | 26-September-<br>2019 | The overall rationale for this amendment is to clarify patient management with regards to treatment regimen and evaluation of encephalopathy and modification of lymphodepleting regimen for older participants, modification of target dose range for NY-ESO transduced cells and changes related to Health Canada requests including updates to both the Encephalopathy (now Immune Effector Cell-Associated Neurotoxicity or ICANS) and the CRS grading and management criteria. |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| None | None | None |

According to GSK standards, Listing of Race (DM9) is required. Due to differences in Adaptimmune data collection, only Listing of Demographic Characteristics (DM2) will be displayed which will include race information.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the safety and tolerability of autologous genetically modified T cells (NY-ESO-1 <sup>c259</sup> T) in human leukocyte antigen (HLA) HLA-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive participants with NY-ESO-1 and/or LAGE-1a positive advanced NSCLC. | <ul> <li>Adverse events (AE), including serious adverse events (SAE);</li> <li>Change of laboratory assessments, including chemistry, hematology, coagulation</li> <li>Cardiac and pulmonary assessments, including electrocardiogram (ECG) and pulmonary function (pulse oximetry);</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of NY-<br>ESO-1 <sup>c259</sup> T | <ul> <li>Investigator-Assessed Overall Response Rate (ORR)</li> <li>Time to response</li> <li>Duration of response</li> <li>Disease Control Rate (DCR)</li> <li>Progression-free Survival (PFS)</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the persistence, phenotype and functionality of NY-ESO-1 <sup>c259</sup> T To understand mechanisms of resistance to NY-ESO-1 <sup>c259</sup> T | <ul> <li>Correlate persistence, phenotype and functionality of NY-ESO-1c259T in the peripheral blood and/or tumor with response to treatment</li> <li>Correlate circulating cytokines with cytokine release syndrome (CRS)</li> <li>Correlate changes in immunosuppressive myeloid cells and Tregs in peripheral blood versus tumor</li> <li>Correlate changes in immunosuppressive myeloid cells and Tregs in peripheral blood and tumor with treatment response</li> <li>Investigate the immune contexture of each participants' tumor over time and to understand mechanisms of tumor resistance, escape and treatment response</li> <li>Determine whether loss of NY-ESO-1c259T expression in tumor is a resistance mechanism</li> </ul> |
| To evaluate antigen spreading as a mechanism of response | Correlate clonal outgrowth of T cell populations with<br>response following T cell infusion |
| To document the exposure and immunogenicity with NY-ESO- 1°259T The exposure the exposure the exposure and immunogenicity with NY-ESO- | Change of anti-NY-ESO-1c259T antibodies |
| To evaluate the survival benefit of<br>NY-ESO-1c259T | Overall Survival (OS) |
| To evaluate the efficacy of NY-<br>ESO-1 <sup>c259</sup> T per immune-related | <ul><li>Overall Response Rate (ORR) per irRECIST</li><li>Time to response (irRECIST)</li></ul> |

# 208749 | Statistical Analysis Plan RAP 02 Oct 2020 | TMF-2069301 | 1.0


| Objectives | Er | ndpoints |
|---|---|---|
| Response Evaluation Criteria in | • | Duration of response (irRECIST) |
| Solid Tumors (irRECIST) | • | Progression-free Survival (PFS, irRECIST) |

### 2.3. Study Design



\*participants, who have a confirmed response (or have stable disease for >4 months) and subsequently have documented PD and whose tumors continue to express NY-ESO-1 as verified by assay performed in biopsied tissue, can be considered for a second infusion with engineered T cells

#### Design Features

- This is a pilot, open-label study of genetically engineered NY-ESO-1<sup>c259</sup>T cells in HLA-A\*02:01, HLA-A\*02:05 and/or HLA-A\*02:06 participants with advanced NSCLC.
   Approximately 10 participants will be enrolled in this study. Sample size was chosen based on clinical judgement and the study is not powered to conduct statistical hypothesis testing.
- Participants will have been screened for the presence HLA-A\*02:01, HLA-A\*02:05 and/or HLA-A\*02:06 and have NY-ESO-1 and/or LAGE-1a expression on the tumor to be eligible to enrol in the study. Prior to the administration of lymphodepleting chemotherapy, participants must have failed at least one prior platinum-containing regimen and have PD. All other eligibility criteria will be reconfirmed and baseline tumor measurements obtained.
- The Screening Phase starts from the time the participant signs the ICF until leukapheresis.
   Eligible participants then enter the Interventional Phase 1 of the study (first T cell infusion) which runs from the day of leukapheresis until progressive disease (PD), death, or followed for 2 years post- T-cell infusion, whichever is shorter
- Following Screening, participants meeting all eligibility criteria will undergo leukapheresis to obtain cells for the manufacture of autologous NY-ESO-1c259 TCR bearing T cells.
- When the NY-ESO-1c259T cells are available, participants will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by infusion of NY-ESO-1c259 transduced T cells in the range of 1 x 10<sup>9</sup> to 6 x 10<sup>9</sup> transduced cells.
- The time point for administration of lymphodepleting chemotherapy and subsequent infusion of NY-ESO-1c259 TCR bearing T cells will be staggered for the first 3 participants enrolled. Participants may receive lymphodepleting chemotherapy as defined in Table 2 (in protocol) only after the previously enrolled participant has had a minimum safety observation period of 21 days following their NY-ESO-1c259 T cell infusion. This 21-day observation period shall remain for the first 3 participants enrolled. If 2 or more participants among the first 3 participants enrolled experience a severe study-related toxicity, enrollment will be paused for evaluation by the Sponsor and Investigators, otherwise, an additional 7 participants will be entered.

208749

| Overview of St | tudy Design and Key Features |
|---|---|
| | <ul> <li>A participant will be considered completing the Interventional Phase 1 of the study when he/she has PD or has died prior to PD, or 2 years after the NY-ESO-1c259T cell infusion, whichever is shorter. A participant will be considered completing the Interventional Phase 2 of the study when he/she has PD, or has died prior to PD, or 6 months after the NY-ESO-1c259T cell infusion, whichever is shorter. All participants completing the Interventional Phase of the study will be rolled over to a long-term follow-up (LTFU) Protocol (GSK208756) for observation of delayed AEs for 15 years post-infusion in accordance Food and Drug Administration (FDA) and European Medicines Agency (EMA) requirements for gene therapy clinical trials.</li> <li>Following the initial infusion, participants, who have a confirmed response (or have stable disease for &gt;4 months) and subsequently have documented PD and whose tumors continue to express NY-ESO-1 and/or LAGE-1a as verified by assay performed in biopsied tissue, can be considered for a second infusion with engineered T cells.</li> </ul> |
| Dosing | <ul> <li>When the NY-ESO-1c259T cells are available, participants will undergo lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by infusion of NY-ESO-1c259 transduced T cells in the range of 1 x 10<sup>9</sup> to 6 x 10<sup>9</sup> transduced cells. The lymphodepleting regimen in this study consists of fludarabine 30mg/m²/day at Days -8, -7, -6 and -5 and cyclophosphamide 900mg/m²/day intravenously at Days -7, -6, and -5.</li> <li>Participants that qualify for a second infusion will receive the same lymphodepleting chemotherapy regimen and T cell infusion as received during the first T cell infusion</li> </ul> |
| Time & | [Refer to Appendix 2: Schedule of Activities] |
| Events | |
| Treatment | This is a single arm open-label unblinded study treated with autologous T cells transduced |
| Assignment | with lentivirus encoding enhanced TCR specific for NY-ESO-1. |
| Interim | No formal interim analyses for efficacy or futility are planned for this study. |
| Analysis | |

## 2.4. Statistical Analyses

The study is not powered to conduct any hypothesis testing on either primary and secondary endpoints. All analyses will be descriptive in nature. Continuous data will be summarized including means, medians, standard deviations, and ranges. Categorical data will be summarized using frequency counts and percentages. Graphical summaries of the data will be presented as appropriate. Time-to-event endpoints will be summarized as the median, and the 25<sup>th</sup> and 75<sup>th</sup> percentiles and displayed graphically using Kaplan-Meier method if data warrant.

#### 3. PLANNED ANALYSES

## 3.1. Primary Analyses

The primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants who have received the first NY-ESO-1<sup>c259</sup>T cell infusion have progressed, or have died, or have been followed for 2 years, or the last participant who has received the second NY-ESO-1<sup>c259</sup>T cell infusion has been followed 6 months after the NY-ESO-1<sup>c259</sup>T cell infusion, progressed, or has died, whichever is later.
- 2. All required database cleaning activities have been completed and database release (DBR) and database freeze (DBF) has been declared by Data Management

If the primary analyses are expected to occur shortly before the final analyses, the study team may decide to conduct only the final analyses.

#### 3.2. Final Analyses

The final analyses will be performed after the completion of the following sequential steps. If the primary analysis and final analysis occurs at the same time, only final analysis will be performed.

- 1. All participants who have received the first NY-ESO-1<sup>c259</sup>T cell infusion have progressed, have died, have been followed 2 year after the first NY-ESO-1<sup>c259</sup>T cell infusion, or have withdrawn from the study; the last participant who has received the second NY-ESO-1<sup>c259</sup>T cell infusion either has been followed until disease progression or withdraws from the study. If LTFU protocol is not available when a participant completes the Interventional Phase, participant can be followed under this protocol until LTFU protocol becomes available. The final analyses will be conducted when all participants are off-study.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants that signed screening informed consent | <ul> <li>Screen Failures</li> </ul> |
| Intent-to-Treat<br>(ITT) | All participants who were enrolled in the trial and met all eligibility criteria | <ul> <li>Primary Study Population </li> <li>Primary Safety</li> <li>Sensitivity Efficacy (ORR and DCR) </li> </ul> |
| Modified Intent-<br>To-Treat (mITT) | All participants in the ITT population who receive NY-<br>ESO-1 <sup>c259</sup> T cell infusion. | Sensitivity Study Population |

208749

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | | <ul> <li>Primary Safety (where appropriate)</li> <li>Sensitivity Safety (where appropriate)</li> <li>Primary Efficacy</li> </ul> |
| Modified Intent-to<br>Treat 2 (mITT2) | All participants that received a second T cell infusion | <ul><li>Efficacy</li><li>Safety</li><li>Study Population</li></ul> |

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarized and all protocol deviations, including both major and minor will be listed.

Protocol deviations will be tracked in accordance with the Protocol Deviation Specification Form by the study team throughout the conduct of the study and sent to Data Manger and Biostatistics Lead in a spreadsheet. There will be no data-driven protocol deviation tracked.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | |
|------------------------------|---|
| Data Displays for Reporting | |
| Description Order in TLF | |
| GSK794 | 1 |

Note that all data displays (Tables, Figures, and Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### 5.2. Baseline Definitions

Unless specified otherwise, baseline measurements should be the most recent value prior to initiating lymphodepletion and should occur within 7 days prior to initiating lymphodepletion. Initiation of lymphodepletion should start on Day -8, but may start on Day -7 if the participant was treated before consenting to Protocol Amendment 2 or after amendment 4 and is  $\geq 60$  years old. If an assessment is not available, then the last assessment prior to that visit would be used even if it occurred more than 7 days prior to initiation lymphodepletion. If time is not collected, assessments taken on the day of lymphodepleting chemotherapy are assumed to be taken prior to lymphodepletion and used as baseline.

For laboratory data, baseline will be defined as the most recent, non-missing value from a central laboratory within 7 days prior to the lymphodepleting chemotherapy. If there are no central labs collected for a participant and a lab test prior to the lymphodepletion, the most recent, non-missing value from a local laboratory within 7 days prior to the lymphodepletion will be defined as the baseline values.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

For participants who did not receive lymphodepleting chemotherapy during the study, baseline will be defined as the latest, non-missing collected value.

For participants that receive a second T-cell infusion, a second baseline associated with second lymphodepletion and infusion will be derived and used for all Second Infusion Phase displays. For all endpoints, except laboratory data, the window for baseline will be <=28 days prior to the initiation of second lymphodepletion chemotherapy, instead of 7 days. For laboratory data (lymphocyte subset (CD3/CD4/CD8), hematology, chemistry, coagulation and urinalysis), baseline will be within 7 days of lymphodepletion as described above for the first infusion.

208749

| Parameter | Study Assessments Considered as Baseline | |
|---|---|---|
| | Screening Informed Consent | Within 7 days prior to initiating lymphodepletion |
| Target and Non-target lesions | | X |
| Hematology,<br>Chemistry, C-reactive<br>protein (CRP), CMV<br>PCR, Additional Lab | | X |
| Vital Signs, Physical Exam, ECOG | | Х |
| Electrocardiograms | | X |
| Cytokines | | X |
| Demography | Х | |

#### 5.3. Multicenter Studies

Data from all participating centers that enrol and treat patients will be pooled prior to analysis.

It is anticipated that participant accrual will be spread thinly across centers and summaries of data by center would be unlikely to be informative and will not, therefore, be provided

## 5.4. Examination of Covariates, Other Strata, and Subgroups

No covariates or strata will be use in analysis and no subgroup analysis will be performed.

# 5.5. Multiple Comparison and Multiplicity

No formal statistical testing will be performed; therefore, no adjustments for multiple comparisons or multiplicity are planned.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices: Note that all data displays (Tables, Figures, and Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

| Section | Component |
|---------|----------------------------------------------------------------|
| 14.3 | Appendix 3: Assessment Windows |
| 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 14.6 | Appendix 6: Derived and Transformed Data |

# 208749 | Statistical Analysis Plan RAP 02 Oct 2020 | TMF-2069301 | 1.0


| Section | Component |
|---------|-----------------------------------------------------|
| 14.7 | Appendix 7: Reporting Standards for Missing Data |
| 14.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the ITT population, unless otherwise specified. The mITT population is the secondary analysis population.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, concomitant medications, disease characteristics at initial diagnosis and at screening, prior and on-study anti-cancer therapy, surgical/medical procedures, substance use, and study treatment exposure will be based on GSK Core and Oncology Data Standards. Study population listings will include second infusion data. Details of the planned displays are presented in Appendix 10: List of Data Displays.

### 6.2. Disposition of Participants

A summary of the number of participants in each of the analysis populations described in Section 4 will be provided. A listing of participants excluded from analysis populations will also be provided.

A summary and listing of screening status and screen failures will be provided using the screened population.

Reason for discontinuation, completion of study, and primary reason for study withdrawal will be summarized in the order they are displayed in the eCRF. Participant status will be displayed with the categories and subcategories Completed study (death, progressive disease, completed 2 years of follow-up), Ongoing or did not complete study with reasons from the CRF. A summary of end of study status for ITT participants will be produced with the reasons Death, Moved to LTFU study, withdrew consent, lost-to-follow-up and death. For participants that are not dosed, end of study reason is equivalent to end of treatment phase reason. Participants dosed and that have a death date in the database are classified with end of study reason=Death. Otherwise, end of treatment phase reason is used as the end of study reason, unless end of treatment phase reason is Progression. If end of treatment phase reason is Progression, then End of Study reasons is not available.

Listing of reasons for study withdrawal for both Interventional Phase 1 and 2 will be provided. A listing of subject status will be generated, including participant number, lymphodepletion, date and dose of T cell infusion, study completion, and date and reason of discontinuation/completion of interventional phase.

#### 6.3. Protocol Deviations

Only important protocol deviations will be summarized and listed and will include inclusion/exclusion deviations as well as other deviations. Protocol deviations will be classified as 'major' and 'minor' based on Protocol Deviation Specifications.

A separate summary and listing of inclusion/exclusion deviations will also be provided

#### 6.4. Demographic and Baseline Characteristics

Disease characteristics at initial diagnosis, time since initial diagnosis in months, stage of lung cancer at initial diagnosis, disease stage at enrolment, and histology will be summarized and listed. In addition to those stated above, date of initial diagnosis will be listed. Refer to Section 14.6.2 for time since initial diagnosis derivation rules.

Disease characteristics at screening, tumor type, anatomical location, number of prior radiotherapy regimens, number of prior systemic therapy regimens, NY-ESO-1 status and HLA status will be summarized and listed. In addition to those stated above, date of blood collection date of biopsy for antigen testing will be listed.

A summary of disease burden at baseline, including number of organs involved and location of disease at baseline, will be produced. Both target and non-target lesions at baseline will be included.

The demographic characteristics at baseline (e.g., race, age, ethnicity, sex, height, body weight, and body mass index (kg/m^2)) will be summarized and listed. Age, height, weight, and bmi will be summarized using the mean, standard deviation, minimum, median and maximum. Age will be summarized by GSK IDSL standard as ≤18, 19-64, ≥65. The count and percentage will be computed for sex and ethnicity. Age at T-cell infusion will be reported for MITT subjects. If date of T-cell infusion is not available, age at study eligibility is reported for ITT subjects.

In a separate summary, age will also be categorized and summarized by 18-64, 65-84 and ≥85 using EudraCT.

Medical conditions will be listed and summarized.

A summary of substance use will be presented, including smoking history, years smoked, and packs per day. A supporting listing will be provided.

# 6.5. Study Treatment Exposure

Number and percentage of participants receiving apheresis procedure, lymphodepleting therapy, and T cell infusion will be summarized for the first T-cell infusion.

A listing of study treatment will be provided, including participant number, total number of transduced cells, percent of cells transduced, T-cell infusion date, study day, start time and end time for first and second T-cell infusion.

The total number of first infusion transduced T cells will be summarized using mean, standard deviation, median and range. Also, the total number of transduced T cells will be categorized into < 1, >=1 to <=8, and >8 (x  $10^9$  cells).

All dose administration data for lymphodepletion, including cyclophosphamide/mesna and fludarabine, will be presented by participant in a data listing for first and second T-cell infusion.

### 6.6. Anti-Cancer Therapy and Surgery

Prior, bridging, and on-study anti-cancer therapy will be coded using GSK Drug coding dictionary. Anti-cancer therapy and cancer-related surgeries will be reported by the three classifications prior, bridging, and on-study, defined in Section 14.4.1.2.

All prior anti-cancer therapy will be summarized by therapy type using the ITT and mITT population. A summary of the number of prior anti-cancer therapy regimens will be provided. Prior anti-cancer surgeries, medications, and therapies will be summarized and anti-cancer therapy, radiotherapy, and surgeries will be listed. Listings of radiotherapy and surgeries will include all procedures that occur before lymphodepletion, and within the listings, bridging procedures will be flagged per Section 14.4.1.2. Prior anti-cancer therapy will be listed and bridging anti-cancer therapy will be provided in a separate listing.

On-study anti-cancer therapies will be summarized using the mITT population. A summary of the number of on-study anti-cancer therapy regimens will be provided. On-study anti-cancer surgeries, medications, and therapies will be summarized, and time from T-cell infusion to first post-treatment anti-cancer therapy will be included. On-study anti-cancer therapy and surgeries will be listed. On-study therapies occurring after second infusion, defined as start date on or after second lymphodepletion chemotherapy, will be flagged in the listings.

Tumor biopsies will be listed.

#### 6.7. Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary, and will be summarized and listed. The summary of concomitant medications will show the number and percentage of participants taking concomitant medication by Ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients. Anatomical Therapeutic Chemical (ATC) classification Level 1 (Body System) information will be included in the dataset created but will not appear on the listing or summary.

In the summary of concomitant medications, each participant is counted once within each unique ingredient. For example, if a participant takes Amoxycillin on two separate occasions, the participant is counted only once under the ingredient 'Amoxycillin'. In the summary of concomitant medications, the ingredients will be summarized by the base only.

Concomitant medications and blood products will also be listed. Concomitant medications and blood products occurring after second infusion, defined as start date on or after second lymphodepletion chemotherapy, will be flagged in the listings.

Definition of concomitant medication study phases are provided in Section 14.4.1.1.

#### 7. EFFICACY ANALYSES

Lesion assessment method and timing, evaluation of disease, disease progression and response criteria for all efficacy analyses will be conducted according to RECIST (version 1.1) [Eisenhauer, 2009].

To be assigned a status of SD, follow-up disease assessment must have met the SD criteria at least once after T-cell infusion at a minimum of 7 weeks (49 days).

If a participant is found to have a tumor response by imaging, a follow-up confirmation scan must be done no earlier than 28 days following the scan when response or disease progression first seen.

Independent review of scans may be performed for participants at the sponsor's discretion. Analysis of independent reviewer data will not be included in the RAP, but may be conducted as an ad hoc exploratory analysis.

Anti-cancer therapy for efficacy censoring includes systemic therapy, radiotherapy, anti-cancer surgery, and tumor biopsy resections.

The efficacy analyses will be based on the mITT population, unless otherwise specified. Both ORR and DCR will also be summarized based on the ITT population. Analysis of ORR will also occur for second infusion efficacy based on the mITT2 population. Second infusion efficacy displays will summarize efficacy on or after second infusion baseline.

# 7.1. Secondary Efficacy Analyses

### 7.1.1. Endpoint / Variables

ORR

Overall Response Rate (ORR) is defined as the percentage of participants with a confirmed PR or CR as the BOR, as assessed by the RECIST 1.1 Criteria.

Best Overall Response (BOR) is defined as the best confirmed response (Complete Response (CR) > Partial Response (PR) > Stable Disease (SD) > Progressive Disease (PD) > Not Evaluable (NE)) from T cell infusion date until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the RECIST 1.1 Criteria.

DCR

Disease Control Rate (DCR), defined as the percentage of participants with a SD or better as the BOR (i.e., Confirmed PR, confirmed CR, or SD  $\geq$  12 weeks, as assessed by the RECIST 1.1 Criteria).

A status of SD durability will be assigned if follow-up disease assessment has met the SD criteria at least once after the first dose at a minimum of 12 weeks.

208749

DOR

Duration of response (DoR), defined as the interval of time in months from first documented evidence of PR or better to the time when disease progression is documented as assessed by the RECIST 1.1, or death due to any cause among participants with a confirmed PR or CR as the BOR. Censoring rule will follow those for PFS as specified in Table 2.

TTR

Time to response (TTR), defined as the interval of time (in months) between the date of T-cell infusion and the first documented evidence of response (PR or CR) in the subset of participants with a confirmed PR or CR as the BOR as assessed by the RECIST 1.1.

PFS

Progression-free survival (PFS), defined as the interval of time (in months) between the date of T-cell infusion and the earlier of the date of disease progression as assessed by the investigator per RECIST 1.1 criteria and the date of death due to any cause. Determination of dates of PFS events and dates for censoring are described in Table 2.

If a participant has neither progressed nor died nor started new anti-cancer therapy, PFS will be censored at the date of the last adequate disease assessment. The acceptable imaging modalities for this study are:

- Diagnostic-quality computerized tomography (CT) scan with oral and/or IV iodinated contrast of the chest and abdomen/pelvis (CT is the preferred modality for tumor assessments):
- Magnetic resonance imaging (MRI) of the abdomen/pelvis acquired before and after gadolinium contrast agent administration and a non-contrast enhanced CT of the chest, if a participant is contraindicated for contrast enhanced CT;
- MRI of the extremities per site standard of care, if clinically indicated;
- Digital photographs of skin lesions including a ruler for estimating the size of the lesion.

For participants who receive subsequent anti-cancer therapy the following rules will apply:

• If anti-cancer therapy is started without documented disease progression or is started prior to documented disease progression, PFS will be censored at the date of the last adequate disease assessment that is no later than the date of initiation of anti-cancer therapy (i.e. if an assessment occurs on the same day as the start of new anti-cancer therapy the assessment will be used, as it will be assumed the assessment occurred prior to the administration of new anti-cancer therapy).

- If a participant has only a baseline visit or does not have an adequate disease assessment that is no later than the date of initiation of subsequent anti-cancer therapy, PFS will be censored at the date of T cell infusion.
- If the start date of the subsequent anti-cancer therapy is partial (i.e. either missing the day but has the month and year available or missing both day and month), the imputation rules described in Section 14.7.2 will be applied. No imputation will be made for completely missing dates.

208749

# Table 2 Assignments of Progression and Censoring Dates for PFS Analysis

| Scenario | Date of Event (Progression/Death) or Censored | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| No baseline assessments <sup>4</sup> and the participant has not died | Day 1 ( NY-ESO-1 <sup>c259</sup> T cell infusion) | Censored |
| No adequate post-baseline assessments before start of new anti-cancer therapy and the participant has not died | Day 1 ( NY-ESO-1 <sup>c259</sup> T cell infusion) | Censored |
| Progression documented between scheduled visits | Date of assessment of progression <sup>1</sup> | Event |
| With adequate post-baseline assessment but no progression (or death) | Date of last 'adequate' assessment of response <sup>2</sup> | Censored |
| With adequate post-baseline assessment and new anticancer treatment started (prior to documented disease progression). <sup>3</sup> | Date of last 'adequate' assessment of response <sup>2</sup> (on or prior to starting anti-cancer therapy) | Censored |
| Death before first scheduled assessment | Date of death | Event |
| Death (regardless of having baseline assessment) before missing two scheduled assessments and no progression | Date of death (Use rule below to determine missing two scheduled assessments) | Event |
| Death (regardless of having baseline assessment) or progression after more than two missed scheduled assessment | Day 1 ( NY-ESO-1 <sup>c259</sup> T cell infusion) if there is no adequate post-baseline assessment or date of last 'adequate' assessment of response (Prior to missed assessments): | Censored |
| | As the assessment schedule changes through the course of the protocol (i.e. every 8 weeks until week 24, then every 3 months from month 9 to month 24, and then every 6 months thereafter), the following rules will be used for identifying extended loss to follow up or extended time without an adequate assessment (i.e. two or more missed assessments). • If PFS event is on or prior to week 24 + 7 days (Day 175), then | |
| | a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment | |

| Scenario | Date of Event (Progression/Death) or Censored | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| | during the time period of 126 days (16 weeks+7 days+7 days) prior to PFS event; | |
| | • Else if PFS event is after week 24 + 7 days (Day 175) and on or prior to the first scheduled disease assessment date (month 9 + 14 days, day 288), then a participant will be identified as an extended loss to follow up if the participant missed both week 16 and week 24 disease assessments: | |
| | o If PFS event is after week day 175 (week 24 + 7 days) and on or prior to day 203 (week 28 + 7 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 126 days (16 weeks+7 days+7 days) prior to PFS event; | |
| | <ul> <li>Else if PFS event is after day 203 (week 28 + 7 days) and on or prior to day 231 (week 32 + 7 days) then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 154 days (20 weeks+7 days + 7 days) prior to PFS event;</li> </ul> | |
| | <ul> <li>Else if PFS event is after day 231 (week 32 + 7 days) and on or prior to day 288 (month 9 + 14 days) then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 183 days (24 weeks+7 days + 7 days) prior to PFS event;</li> </ul> | |
| | • Else if PFS event is after day 288 (month 9 + 14 days) and on or prior to the second scheduled disease assessment date (month | |

| Scenario | Date of Event (Progression/Death) or Censored | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| | 12 + 14 days, day 379), then a participant will be identified as an extended loss to follow up if the participant missed both week 24 and month 9 disease assessments: | |
| | o If PFS event is after day 288 (month 9 + 14 days) and on or prior to day 318 (month 10 + 14 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 168 days (8 weeks + 3 months+7 days + 14 days) prior to PFS event; | |
| | <ul> <li>Else if PFS event is day 318 (month 10 + 14 days) and on or prior to day 349 (month 11 + 14 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 199 days (8 weeks + 4 months+7 days + 14 days) prior to PFS event;</li> </ul> | |
| | <ul> <li>Else if PFS event is after day 349 (month 11 + 14 days) and on or prior to day 379 (month 12 + 14 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 219 days ((9mon-24 weeks=106 days) + 3 months +7 days + 14 days) prior to PFS event;</li> </ul> | |
| | • Else if PFS event is after day 379 (month 12 + 14 days) and on or prior to day 745 (month 24 + 14 days), then a participant will be identified as an extended loss to follow up if the participant | |

| Scenario | Date of Event (Progression/Death) or Censored | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| | did not have an adequate disease assessment during the time period of 211 days (6 months+14 days + 14 days); | |
| | • Else if PFS event is after day 745 (month 24 + 14 days) then a participant will be identified as an extended loss to follow up if they missed 1 visit | |
| | <ul> <li>Else if PFS event is day 745 (month 24 + 14 days) and on or prior to day 776 (month 27 + 14 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 211 days (6 months + 14 days + 14 days) prior to PFS event;</li> </ul> | |
| | <ul> <li>Else if PFS event is after day 776 (month 27 + 14 days), then a participant will be identified as an extended loss to follow up if the participant did not have an adequate disease assessment during the time period of 274 days (6 months + 3 months) prior to PFS event;</li> </ul> | |
| | PFS will be censored at the date of last adequate disease assessment of response or Day 1, whatever is later, prior to PD/death. | |

The earliest of (i) Date of radiological assessment showing new lesion (if progression is based on new lesion); or (ii) Date of radiological assessment showing unequivocal progression in non-target lesions, or (iii) Date of last radiological assessment of measured lesions (if progression is based on increase in sum of measured lesions)

<sup>&</sup>lt;sup>2</sup> An adequate assessment is defined as an assessment where the Investigator determined response is CR, PR, or SD.

<sup>&</sup>lt;sup>3</sup> If PD and New anti-cancer therapy occur on the same day assume the progression was documented first e.g., outcome is progression and the date is the date of the assessment of progression).

<sup>&</sup>lt;sup>4</sup> No baseline assessment defined as baseline scan performed outside of the protocol defined window (>7 days before start of lymphodepletion) or no baseline scan at all.

208749

#### 7.1.2. Summary Measure

ORR

The number and percentage of participants with the BOR in the following response categories will be summarized: CR, PR, SD, PD, NE and overall response (CR+PR), The exact 95% CI for ORR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of response. ORR will be summarized for the ITT, mITT, and mITT2 population.

Change in target lesions from baseline over time will be shown in a spider plot. A waterfall plot showing the maximum percent reduction from baseline in tumor measurement will be also produced.

ORR will be listed.

DCR

The number and percentage of participants with the BOR in the following response categories will be summarized: Confirmed CR, PR, or SD  $\geq$  12 weeks, clinical benefit response (Confirmed CR+PR+SD  $\geq$  12 weeks), PD and NE. The corresponding exact 95% CI for DCR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of DCR. DCR will be summarized for the ITT and mITT population.

DOR

If there are sufficient number of responses at time of primary or final analysis, distribution of DOR will be summarized using the Kaplan-Meier method. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of DOR will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method [Brookmeyer, 1982].

TTR

If there are sufficient number of responses at time of primary or final analysis, time to response at will be summarized descriptively using median, min, max and quartiles in the subset of participants with a confirmed response of PR or CR as the BOR.

PFS

The distribution of PFS will be estimated using the Kaplan-Meier method if data warrant. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of PFS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method [Brookmeyer, 1982].

208749

For DOR and PFS, Kaplan-Meier quantiles along with two-sided 95% CIs will be listed and summarized in months if data warrant. A Kaplan-Meier curve will be produced with 95% confidence bands, if data warrant.

#### 7.1.3. Population of Interest

The secondary efficacy analyses will be based on the mITT population. The ITT is the sensitivity analysis population for Disease Control Rate (DCR) and ORR. If the mITT and ITT populations are identical, only results associated with the mITT population will be reported.

#### 7.1.4. Strategy for Intercurrent Events

For ORR, participants who are not evaluable or have missing response will be treated as non-responders; i.e. they will be included in the denominator when calculating the percentage

For PFS and DOR:

Intercurrent events, such as use of protocol prohibited medication, switching to a different treatment, or withdrawal of consent, are expected. Refer to Table 2 for censoring rules and intercurrent event strategy.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.2. Exploratory Efficacy Analyses

The only exploratory efficacy endpoint that will be reported is overall survival (OS). Endpoints per irRECIST will not be reported.

#### 7.2.1. Overall Survival

Overall Survival (OS), defined as the interval of time (in months) from T-cell infusion to the date of death due to any cause. For participants who have not died at the time of analysis they will be treated as censored and the last date of known contact derived per Section 14.6.3.

#### 7.2.2. Summary Measure

The distribution of OS will be estimated using the Kaplan-Meier method if data warrant. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of OS will be estimated and corresponding two-sided 95% confidence intervals will be estimated using the Brookmeyer-Crowley method [Brookmeyer, 1982].

Kaplan-Meier quantiles along with two-sided 95% CIs will be listed and summarized in months if data warrant. A Kaplan-Meier curve will be produced with 95% confidence bands, if data warrant.

#### 7.2.3. Population of Interest

The exploratory efficacy analyses will be based on the mITT population.

#### 7.2.4. Strategy for Intercurrent Events

Intercurrent events, such as use of protocol prohibited medication, switching to a different treatment, or withdrawal of consent, are expected. If a participant has an intercurrent event that precludes observation of the endpoint death, the patient will be censored at the date of last contact. If the patient has an intercurrent even that does not preclude the observation of the endpoint death, the patient's event will be included in the analysis and the intercurrent event will not be accounted for.

#### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Intent-To-Treat population except for displays that are treatment dependent. In those cases, the modified Intent-To-Treat population will be the primary safety, as detailed in Appendix 10: List of Data Displays. The mITT is the secondary analysis population.

### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. Details on treatment emergent AEs are provided in Section 14.4.2. The details of the planned displays are provided in Appendix 10: List of Data Displays.

AEs will be graded by the investigator according to the National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) v4.03. AEs will be coded to the Preferred Term (PT) level using the Medical Dictionary for Regulatory Affairs (MedDRA) V23.0. Per Protocol V4 effective 26-Sept-2019, CRS events are graded using the American Society for Transplantation and Cellular Therapy grading system [Lee, 2019]. Previous versions of the protocol collected CRS events graded using 2014 criteria [Lee, 2014].

Per the request of the clinical team, various Preferred Terms were combined and will be reported together as one term. The combined terms for MedDRA Version 23.0 are listed in Appendix 12: Combined Preferred Terms. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional combined terms, therefore the list of combined preferred terms will be based on the safety review team (SRT) agreements in place at the time of reporting. Tables that summarize AEs by SOC and PT will use MedDRA preferred terms, as well as any adverse event tables required for disclosure. Most other AE tables will summarized AEs by the combined terms in Appendix 12: Combined Preferred Terms, as detailed in the programming notes in Appendix 10: List of Data Displays.

Tables will summarize all AEs for the ITT population and Treatment Emergent AEs for the mITT population.

A summary of non-serious AEs that occurred in strictly 5% of the participants or above will be provided (no rounding for the percentage will be used in terms of 5% threshold, e.g. events with 4.9% incidence rate should not be included in this table). This summary will contain the number and percentage of participants and the number of occurrences of common non-serious adverse events. The summary table will be displayed by System Organ Class (SOC) and Preferred Term (PT).

A summary of number and percentage of participants with any AEs by maximum grade will be produced. AEs will be sorted by PT in descending order of total incidence. The summary will use the following algorithms for counting the participant:

- **Preferred term row**: Participants experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- **Any event row**: Each participant with at least one AE will be counted only once at the maximum grade no matter how many events they have.

In addition, the frequency and percentage of AEs (all grades) will be summarized and displayed in descending order of total incidence by SOC and PT. In the SOC row, the number of participants with multiple events under the same system organ class will be counted once.

Three separate summaries will be provided for the study treatment related AEs displays. One table will be produced for each of the following: Lymphodepletion-related, T-cell related, and Any Study Treatment-related. A study treatment-related AE is defined as an AE for which the investigator classifies the relationship to study treatment as "Yes", which includes "Definitely Related", "Probably Related" or "Possibly Related". A worst-case scenario approach will be taken to handle missing relatedness data, i.e. the summary table will include events with the relationship to study treatment as 'Yes' or missing. The summary tables by maximum grade will be displayed in descending order of total incidence by PT only.

Second infusion adverse events are defined in Section 14.4.2 and will be identified with a flag in AE listings.

A listing of delayed AEs as-adjudicated by GSK will be provided. GSK adjudicated AEs will be provided as an additional data source.

All AEs will be listed. Additionally, a listing of participant IDs for each individual AE will be produced. Time from second T-cell infusion, Study Day 2, will be included in listings that list data Post-Second Infusion. Study Day 2 is defined in Section 14.6.1

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event including use of all SMQs where applicable. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. A focused and a comprehensive list of MedDRA terms was developed to identify the following AESIs. The details of the planned displays are provided in Appendix 10: List of Data Displays.

The events of special interest include the following categories

- Graft versus host disease
- Guillain-Barre syndrome
- Haematopoietic cytopenias (including pancytopenia and aplastic anaemia)
- Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS)

208749

- Cytokine release syndrome
- Pneumonitis

AESI tables will be reported for the mITT population. All tables below will be summarized using the focused list for all AESI and for the Haematopoietic cytopenia AESI using both the comprehensive and focused list of preferred terms.

For each AESI, time from T cell infusion to first onset (in days) and duration of first occurrence and last occurrence will be summarized for all AESIs.

The number and percentage of participants with these events will be summarized by categories of AESI and preferred term in one table. The summary of event characteristics for each category of AESI will also be provided, including number of participants with any event, number of events, number of participants with any event that is serious, number of participants with any event that is related to study treatment, the outcome of the event, maximum grade and the action taken for the event. The percentage will be calculated in two ways, one with number of participants with event as the denominator and the other with total number of participants as the denominator. The worst-case approach will be applied at participant level for the event outcome and maximum grade, i.e. a participant will only be counted once as the worst-case from all the events experienced by the participant. For action taken to an event, participant will be counted once under each action.

A summary of onset and duration of the first occurrence and last occurrence of all AESIs will be created for each AESI separately. A summary of time to resolution will also be created for each AESI separately. The time to resolution displays summarizes participants with an AESI occurring before study day 28. Among all AESIs occurring before study day 28, the worst-case study day of resolution will be summarized. Additionally, the worst-case AESI duration of all recurrent AESIs will be summarized. Recurrent AESI is defined as additional occurrences of AESIs after initial occurrence before study day 28. Duration is defined as end date-start date+1.

Characteristics, Onset and Duration, and Time to Resolution summaries will not be created if there are 0 or 1 AESI.

# 8.2.1. Cytokine Release Syndrome (CRS) and Graft versus Host Disease (GvHD)

Refer to Section 8.5 and Section 8.6 of the Protocol for the definitions and the grading of CRS and GvHD. Listing for participants experiencing AE of GVHD will be provided, which will include leukapheresis date, chemo start date, T cell infusion date, AE start date, time since infusion (days), AE end date, SAE code, severity, relationship to T cell infusion, and outcome of event. Listing for participants experiencing AE of CRS will also include time from infusion to first CRS (days) and time from infusion to max CRS (days). If data warrant, time from infusion to first occurrence and duration of CRS (days) will be summarized using mean, standard deviation, median, and range. The mock-up shells are in Appendix 11: Example Mock Shells for Data Displays.

#### 8.3. Deaths and Serious Adverse Events

In the event that a participant has withdrawn consent, no data after the withdrawal of consent date from this participant including death is supposed to appear in the database, which should be part of the data cleaning process. All deaths will be summarized based on the number and percentage of participants. This summary will classify participants by time of death relative to the date of T cell infusion as a categorical (>30 days or  $\leq$ 30 days) and primary cause of death (disease under study, treatment related toxicity, or other). A supportive listing will be generated to provide participant-specific details on participants who died.

All SAEs will be tabulated based on the number and percentage of participants who experienced the event. Summaries will be displayed by System Organ Class (SOC) and Preferred Term (PT). Another table will summarize the frequency and percentage of fatal AEs in descending order of total incidence by PT only.

Three separate summaries will be provided for the study treatment related SAEs displays. One table will be produced for each of the following: Lymphodepletion-related, T-cell related, and Any Study Treatment-related. These three summaries will also be reported for Fatal Adverse Events if there are at least 5 participants with fatal study treatment-related AEs. A study treatment-related SAE is defined as an SAE for which the investigator classifies the relationship to study treatment as "Yes", which includes "Definitely Related", "Probably Related" or "Possibly Related". A worst-case scenario approach will be taken to handle missing data, i.e. the summary table will include events with the relationship to study treatment as 'Yes' or missing.

SAEs are included in the listing of all adverse events. Separate supportive listings with participant-level details will be generated for

- Fatal SAEs
- Non-fatal SAEs.

A plot of study duration including study days of any SAE, death, progression, and response will be produced.

# 8.4. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

| Clinical Chemistry: | Calcium |
|---|---|
| | Phosphorus |
| | Magnesium |
| | Albumin |
| | Bilirubin |
| | Alanine aminotransferase |
| | Aspartate aminotransferase |
| | Alkaline phosphatase |
| | Lactic acid dehydrogenase |
| | Sodium |
| | Potassium |
| | Bicarbonate |
| | Creatinine* |
| | Chloride |
| | Glucose |
| | Urea |
| | * In participants <65 years of age creatinine clearance will be calculated using the Cockcroft-Gault Method: |
| | *Participants ≥65 years of age must have renal function measured either by 24-hour urine creatinine collection or by nuclear medicine EDTA GFR measurement, according to standard practice at the treating institution. |
| Coagulation Screen: | Prothrombin time or International Normalized Ratio |
| | Activated partial tissue thromboplastin time |
| ECG Parameters: | Heart Rate |
| | Heart Rhythm |
| | PR Interval |
| | RR Interval |
| | QRS Interval |
| | QTc Interval (Fridericia's or Bazett's correction) |

208749

| Hematology: | Red cell count |
|---|---|
| | Hemoglobin |
| | Hematocrit |
| | Mean cell volume |
| | Mean corpuscular hemoglobin |
| | Mean corpuscular hemoglobin concentration |
| | Platelet count |
| | White blood cell count & differential count (percent & absolute) |
| Lymphocyte subset | Absolute cell count and percentage of CD3, CD4, and CD8 |
| Pregnancy Test: | Serum beta-HCG or Urine test |
| Thyroid Function Tests: | TSH with reflex free T4 |
| Urinalysis: | Glucose |
| | Ketones |
| | Specific gravity |
| | Protein |
| | Blood |
| | Microscopy |
| | Bilirubin |
| | pH |
| Infectious disease markers: | HIV 1+2 antibody |
| | Hepatitis B core antibody – if positive, test for HBV DNA |
| | Hepatitis C antibody – if positive, test for HCV RNA |
| | HTLV 1+2 IgG |
| | CMV IgG / DNA PCR |
| | Epstein-Barr virus (EBV) (EBNA) |
| | Syphilis (spirochaete bacterium) rapid plasma regain |
| Other Tests: | Uric Acid |
| | C-reactive protein |

Laboratory grades will be reported using the CTCAE v4.03.

Summary of the post-baseline change of lab values for each visit (including cytomegalovirus (CMV) by polymerase chain reaction (PCR), and C-reactive protein
208749

(CRP)) using mean, median, standard deviation, minimum, and maximum will be provided. Labs that do not have post-baseline values will not be included in the table.

Summaries of worst case grade increase from baseline grade will be provided for all the lab tests that are gradable by CTCAE v4.03. These summaries will display the number and percentage of participants with a maximum post-baseline grade increasing from their baseline grade. Missing baseline grade will be assumed as grade 0. For laboratory tests that are graded for both low and high values, summaries will be done separately and labeled by direction, e.g. sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by CTCAE v4.03, summaries of worst-case changes from baseline with respect to normal range will be generated. The worst case will be chosen from all available tests, including scheduled and unscheduled visits. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized for the worst case post-baseline. If a participant has a decrease to low and an increase to high during the same time interval, then the participant is counted in both the "Decrease to Low" categories and the "Increase to High" categories.

Separate summary tables for hematology, chemistry, urinalysis, and other laboratory tests will be produced. Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of participants with non-missing value at each particular visit.

A supporting listing of laboratory data for participants with any value outside normal range or any value of potential clinical importance will be provided. All laboratory values, including pre-baseline values, will be included in the listing. A separate listing of laboratory data with character values will also be provided.

Detailed derivation of baseline assessment is specified in Section 5.2.

Second infusion lab assessments will be excluded from "worst-case post baseline" in tables. Lab tables will only summarize first-infusion lab values. First infusion displays will summarize lab assessments before second infusion baseline. All listings will include first infusion and second infusion assessments.

#### 8.4.1. Analyses of Liver Function Tests (LFT)

Summaries of hepatobiliary laboratory events including possible Hy's law cases will be provided.

Possible Hy's law cases are defined as any elevated (ALT≥3×ULN and total bilirubin≥2×ULN (with direct bilirubin ≥35% of total bilirubin, if direct bilirubin is measured)) **OR** (ALT≥3×ULN and INR >1.5, if INR is measured). Note that INR measurement is not required and the threshold value stated will not apply to participants receiving anticoagulants.

A scatter plot of maximum total bilirubin versus maximum ALT will be generated. Also a scatter plot of maximum vs baseline for ALT will be produced. Both plots will be produced for first infusion only.

### 8.5. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs, pregnancies, and vital signs will be based on GSK Core Data Standards, unless otherwise specified. Performance status will be summarized and listed based on GSK Oncology Data Standard. The details of the planned displays are presented in Appendix 10: List of Data Displays.

Second infusion assessments will be excluded from "worst-case post baseline" in tables. Tables will be produced for first infusion only. First infusion displays will summarize safety assessments before second infusion baseline. All listings will include first infusion and second infusion assessments.

#### 8.5.1. Performance Status

ECOG performance status will be summarized at baseline and last-assessment for first infusion. Summaries will use frequency and percentage of participants at each planned assessment time. A summary of change from baseline by scheduled visits will be performed, as well as the worst case post-baseline and the best case post-baseline changes during the study (improved, no change, deteriorated).

A supporting listing will also be provided that includes both first infusion and second infusion visits

#### 8.5.2. ECG

A summary of the number and percentage of participants who had normal and abnormal (clinically significant and not clinically significant) ECG findings will be displayed by scheduled visits as well as for the worst case post-baseline. The worst case will be chosen from all available ECG findings, including scheduled and unscheduled visits.

A summary of change from baseline in ECG values will be produced. QtcB and QtcF will be summarized separately.

The number of participants with maximum QTc values (i.e., worst case) post-baseline relative to baseline will be summarized by test (e.g., QTcF Interval, Aggregate) and category. Also, a summary by a categorization of participants' maximum increase (i.e., worst case) in QTc value (e.g., QTcF Interval, Aggregate) post-baseline relative to baseline will be produced. Both QTcB and QTcF are collected, and will be summarized separately.

Listings of abnormal ECG findings and a listing of ECG values of PCI will be provided.

#### 8.5.3. Vital Signs

A summary of change from baseline in vital signs will be provided. Also, a summary of worst case vital signs results by CTCAE criteria and normal range post-baseline relative to baseline will be generated.

A listing of all vital signs data for participants with any value of PCI will be provided. Also there will be a listing of vital signs of PCI.

### 8.5.4. Pregnancies

Pregnancy (or pregnancy of a male participant's partner) is not considered an AE/SAE unless there is reason to believe that the pregnancy may be the result of failure of the contraceptive being used due to interaction with the study drug. However, the investigator shall report all pregnancies immediately to the Sponsor. If participants or participants' partner become pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

## 8.5.5. Replication Competent Lentivirus (RCL) and Persistence of NY-ESO-1<sup>c259</sup>T

The proportion of participants showing >1% gene marked PBMCs one year post-first infusion or one year post-second infusion will be summarized. Only persistence measurements collected before occurrence of second infusion will be considered for one year post-first infusion derivation.

For any patient who has greater than 1% gene marked PBMCs at at least 1 year or beyond post-infusion, integration site analysis will be performed on PBMCs to assess clonality and possible insertional oncogenesis. The proportion of participants who are RCL positive will also be summarized, if data warrant.

The proportion of participants who are RCL positive will also be summarized for all infusions.

RCL results will also be presented in a data listing.

#### 9. BIOMARKER ANALYSES

## 9.1. Exploratory Biomarker Analyses

## 9.1.1. Endpoint / Variables

Persistence, cytokines, and immunohistochemistry data described in this RAP will be reported if data warrant. Any additional exploratory biomarker, including anti-NY-ESO antibodies, and persistence analyses will not be included in this RAP, but may be described in a separate RAP and included in the CSR if data warrant.

## 9.1.2. Summary Measure

#### 9.1.2.1. Persistence of NY-ESO-1<sup>c259</sup>T

Spider plots will be used to graphically summarize persistence (copies/µg DNA) over time for each participant by responders and non-responders for first infusion and second infusion separately. Maximum persistence during the study and time to maximum persistence will be summarized overall and for responders and non-responders using descriptive statistics and boxplots for first infusion. If the reported result is Negative, then the value 0 will be used for values deemed < lower limit of quantitation or > upper limit of quantitation, and upper limit of quantitation values will be used for values deemed < lower limit of quantitation or > upper limit of quantitation.

The following calculations will be performed:

copies/cell is calculated with the following formula:

copies/cell=(copies/µg)x(0.0000063 µg DNA/cell)

Percent gene marked peripheral blood mononuclear cells (PBMCs) =(copies/cell) \*100

The final reported result of copies/µg DNA is calculated as follows:

copies/µg DNA=copies per well/µg DNA per well

A listing of persistence will be provided and will include coefficient of variation, number of positive replicates, copies/cell, copies/DNA, percent gene marked PBMCs (%), detectable result and time to loss of 25%/50%/75% peak persistence, and duration of detectable persistence. Time to loss of 25% of peak persistence will be calculated as the time since T-cell infusion corresponding to observing at least 25% loss of peak persistence. If time to 25% loss of peak persistence is not observed, the last observed time is reported with a "+" appended to the numerical result. The same procedure will be followed for 50% and 75%. Duration of detectable persistence is derived as time from T-cell infusion until persistence is no longer detectable (persistence falls below the detection limit and interpretive result is "Negative"). If persistence remains detectable for the given participant on study, the last observed time is reported with a "+" appended to the numerical result. Peak persistence, duration of detectable persistence and time to loss

of peak persistence will be derived separately for second infusion and presented in the listing.

First infusion figures and tables will summarize persistence collected before second infusion baseline and second infusion figures will summarize persistence on or after second infusion baseline.

#### **9.1.2.2.** Cytokines

If data warrant, boxplots of the maximum post-baseline value and spider plots for select cytokines including but not limited to IL-1 $\beta$ , IL-10, IL-6, TNF- $\alpha$ , and IFN- $\gamma$  will be provided for participants with none or non-serious CRS vs. serious CRS for the overall cohort and for responders vs. non-responders if data warrant. Boxplots and spider plots by responders vs. non-responders will also be created for cytokines IL-7 and IL-15. One spider plot and boxplot will be presented per cytokine.

Cytokine results will be presented by participant in a data listing if data warrant. Prebaseline cytokines will also be included in the listing. Participants with an adverse event of serious CRS will be flagged in the listing. If the reported result is "Fail QC" or "CV>25%", then the value will be set to missing for values deemed < lower limit of quantitation or > upper limit of quantitation. If the reported result is "<LLOQ (ex. <0.25)", the laboratory specified lower limit of quantification/3 will be used. If the reported result is ">ULOQ (ex >2.5)", the laboratory specified upper limit of quantification will be used. If there are multiple baseline values, the value analyzed first will be used as the baseline value

Only cytokine associated with first infusion will be plotted.

#### 9.1.3. Population of Interest

The primary biomarker analyses will be based on the mITT population, unless otherwise specified.

#### 10. PHARMAKOKINETIC ANALYSES

N/A

# 11. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

N/A

208749

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

N/A

208749

## 13. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. *Biometrics*. 1982;38:29-41.

Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). *European Journal of Cancer*. 2009;45(2):228-247.

Lee DW, Gardner R. Current concepts in the diagnosis and management of cytokine release syndrome. *Blood.* 2014;124(2):188-195.

Lee DW, Santomasso BD, Locke FL. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. *Biology of Blood and Marrow Transplantation*. 2019;25:625-38.

208749

## 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Specification document.

208749

## 14.2. Appendix 2: Schedule of Activities

## 14.2.1. Protocol Defined Schedule of Events Interventional Phase I

## Table 3 Schedule of Procedure (Interventional Phase 1)

| | | In | terventi | onal | Phase | 1 | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Leuka-<br>pheresis | Base-<br>line | | phode<br>mother | | | T-cell<br>in-<br>fusion <sup>3</sup> | | t-T-0 | ell Iı | ıfusi | ion | | | | | | | | | | | | | | Comp |
| Day (D) / Week<br>(W) | - 28 D <sup>4</sup><br>of<br>Leuka-<br>pheresis | | D -14<br>to -9 | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D 2 | D 3 | D 4 | D 5 | D 8 | W 2 | 2W 3 | 3 W 4 | 1 W 5 | 6 | W8 | W<br>10 | W<br>1<br>2 | W<br>1<br>6 | W<br>20 | W<br>24 | Every 3<br>Mos<br>Until Yr<br>2. | Every 6<br>Mos<br>Thereafter | etion/<br>Withd |
| Visit Window | | n/a | n/a | n/a | n/a | n/ a | n/a | n/a | ±1 d | lay | • | • | | ±3 ( | lays | • | • | • | ±7 d | ays | | | | | ±14<br>days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 1<br>8 | 19 | 20 | 2<br>1 | 2 | 23 | 24 | 25-30 | 31+ | |
| Clinical As | sessments | and Pro | cedures | 6 (ref | fer to S | Sectio | n 7.4 i | in the Pr | otoco | ol fo | r deta | ails) | | | | | | | | | | | | | | | |
| Informed<br>Consent <sup>7</sup> | X <sub>EDC</sub> | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Demographics | XEDC | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Inclusion/<br>Exclusion | 8<br>Xedc | | X <sup>9</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical<br>History10, and<br>Tobacco Use | X | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical Exam | X | | X | | | | | X | | | | | X | X | | | | | | | | | | X | X | X | |
| Prior/Concomitant Medications11 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECOG | X | | X | | | | | X | | | | | X | X | X | X | | X | X | | X | X | | X | X | X | X |
| Vital Signs /<br>Height/ Weight12 | X | | X | | | | | X13 | X | X | X | X | X | X | | | | | | | | | | | | | X |
| ECG | X | | X | | | | | X | | | X | | X | | | | | | | | | | | | | | |

| | ~ | In | terventi | onal | Phase | 1 | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen-<br>ing<br>Phase <sup>1</sup> | Leuka-<br>pheresis | | - | phode<br>nother | _ | _ | T-cell<br>in-<br>fusion <sup>3</sup> | | t-T-c | ell Iı | ıfus | ion | | | | | | | | | | | | | | |
| Day (D) / Week<br>(W) | - 28 D <sup>4</sup><br>of<br>Leuka-<br>pheresis | | D -14<br>to -9 | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D 2 | D 3 | D 4 | D 5 | D 8 | W<br>2 | W 3 | W 4 | W 5 | 5 W<br>6 | W8 | W<br>10 | W<br>1<br>2 | W<br>1<br>6 | W<br>20 | W<br>24 | Every 3<br>Mos<br>Until Yr<br>2. | Every 6<br>Mos<br>Thereafter | Compl<br>etion/<br>Withd<br>rawal <sup>5</sup> |
| Visit Window | | n/a | n/a | n/a | n/a | n/ a | n/a | n/a | ±1 d | lay | I. | <u> </u> | | ±3 ( | days | <u> </u> | 1 | <u> </u> | ±7 d | ays | <u> </u> | 1 | | <u>I</u> | ±14<br>days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 1<br>8 | 19 | 20 | 2<br>1 | 2 2 | 23 | 24 | 25-30 | 31+ | |
| ECHO/MUGA | 4<br>X <sub>EDC</sub> | | | | | | | | | | | | | | | | | | | | | | | | | | |
| CT / MRI <sup>14</sup> | X <b>4</b> | | X | | | | | | | | | | | | | | | | X | | | X | | X | X | X | X |
| Brain MRI <sup>28</sup> | X | | X | | | | | See foo | tnote | 28 | | | | | | | | | | • | , | | | | • | • | • |
| ICE <sup>29</sup> | | | | | | | | See foo | tnote | 29 | | | | | | | | | | | | | | | | | |
| Chest X-ray | | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| PFTs15 | X <sub>EDC</sub> | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Lymphocyte<br>Subset<br>(CD3/CD4/CD8) | XEDC | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hematology | 4<br>Xedc | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Chemistry | X <b>4</b> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | | X | X | | X | X | X | X |
| Coagulation Tests | X4 | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test16 | X | | X | | | | | X | | | | | | | | X | | | X | | X | X | X | X | X | X | X |
| Urinalysis | X4 | | X | | | | | | | | | | | | | | | | | | T | | | | | | |
| Infectious disease markers <sup>17</sup> | XEDC | | | | | | | | | | | | | | | | | | | | | | | | | | |

| | ~ | In | terventi | onal l | Phase | 1 | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen-<br>ing<br>Phase <sup>1</sup> | Leuka-<br>pheresis | Base-<br>line | | phode<br>mother | | | T-cell<br>in-<br>fusion <sup>3</sup> | Post | :-Т-с | ell I | nfusi | ion | | | | | | | | | | | | | | Comp |
| Day (D) / Week<br>(W) | - 28 D <sup>4</sup><br>of<br>Leuka-<br>pheresis | | D -14<br>to -9 | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | | | D 3 | D 4 | D 5 | D 8 | W<br>2 | W 3 | 3 W 4 | 1 W 5 | 6 W | W8 | W<br>10 | W<br>1<br>2 | W<br>1<br>6 | W<br>20 | W<br>24 | Every 3<br>Mos<br>Until Yr<br>2. | Every 6<br>Mos<br>Thereafter | etion/<br>Withd |
| Visit Window | | n/a | n/a | n/a | n/a | n/ a | n/a | n/a | ±1 d | lay | <u> </u> | | 1 | ±3 ( | days | | 1 | 1 | ±7 d | ays | | 1 | | | ±14<br>days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 1 | 19 | 20 | 2 | 2 2 | 23 | 24 | 25-30 | 31+ | |
| CMV IgG and PCR <sup>18</sup> | | | X | | | | | X | | | | | | X | | X | | X | X | | | | | | | | |
| TSH with free T419 | | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| CRP <sup>20</sup> | | | X | | | | | X | | | X | | X | X | | X | | | | | | | | | | | |
| Uric acid | | | X | | | | | X | | | | | | | | | | | , | | | | | | | | |
| GFR or 24h<br>urine <b>21</b> | X | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Events <sup>22</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vector Copies<br>(Persistence for<br>Safety) <sup>23</sup> | | | | | | | | X | | | | | | | | | | | | | X | | | X | X23 | X23 | |
| VSV-G DNA<br>(RCL) <sup>24</sup> | | | | | | | | X | | | | | | | | | | | | | X | | | X | X24 | X24 | |
| Leukapher | esis, Lym | phodeple | ting Ch | emot | herapy | & I1 | ovestig | ational l | Prod | uct A | Adm | inist | ratio | n | | | 1 | | • | | ı | 1 | | • | 1 | | <u>4</u> |
| Leukapheresis | | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Fludarabine | | | | X | X | X | X | | | | | | | | | | | | | | | | | | | | |

| | C | In | terventi | onal 1 | Phase | 1 | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen-<br>ing<br>Phase <sup>1</sup> | Leuka-<br>pheresis | Base-<br>line | | phode<br>nother | | 2 | T-cell<br>in-<br>fusion <sup>3</sup> | | t-T-c | ell Iı | ıfusi | on | | | | | | | | | | | | | | Compl |
| Day (D) / Week<br>(W) | - 28 D <sup>4</sup><br>of<br>Leuka-<br>pheresis | | D -14<br>to -9 | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D 2 | D 3 | D 4 | D 5 | D 8 | W<br>2 | W 3 | W 4 | W 5 | 6 | W8 | W<br>10 | W<br>1<br>2 | W<br>1<br>6 | W<br>20 | W<br>24 | Every 3<br>Mos<br>Until Yr<br>2. | _ | etion/<br>Withd |
| Visit Window | | n/a | n/a | n/a | n/a | n/ a | n/a | n/a | ±1 ( | lay | | | | ±3 ( | lays | | <u> </u> | | ±7 d | ays | | | | 1 | ±14<br>days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 1 | 19 | 20 | 2 | 2 2 | 23 | 24 | - | 31+ | |
| Cyclophos-<br>phamide | | | | | X | X | X | | | | | | | | | | | | | | | | | | | | |
| NY-ESO-1 <sup>c259</sup> T | | | | | | | | X | | | | | | | | | | | | | | | | | | | |
| Correlative | Studies a | and Resea | arch As | sessm | ents (r | refer | to Sec | tion 7.5 i | n th | e pro | toco | l for | deta | ils) | | 1 | | 1 | 1 | 1 | 1 | 1 | | | | <u> </u> | |
| Pharmacogenetic analysis | | | X <sup>25</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Tumor biopsy <sup>26</sup> | | | <b>X</b> 26a | | | | | | | | | | | | | | | | X | | | | | | | | X |
| Liquid biopsy <sup>26b</sup> | | | X | | | | | | | | | | | | | | | | X | | | | | | | | X |
| Cell phenotype<br>and Functional<br>Assays, | | | X | | | | | X | | | X | | X | X | | X | | | X | | X | | | | | | X |
| Cytokine<br>Analyses <sup>20</sup><br>& Humoral Anti-<br>Infused Cell<br>Responses | | | X | | | | | <sub>X</sub> 27 | Х | X | X | X | X | X | X | X | | | X <sup>2</sup> 7 | | X | | | | | | X |

208749

| | ~ | Int | terventi | onal l | Phase 1 | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ina | Leuka-<br>pheresis | | | phodep<br>nothera | _ | | T-cell<br>in-<br>fusion <sup>3</sup> | Post | t-T-c | ell I | nfus | ion | | | | | | | | | | | | | | Compl<br>etion/ |
| Day (D) / Week<br>(W) | - 28 D <sup>4</sup><br>of<br>Leuka-<br>pheresis | | D -14<br>to -9 | | l . | D<br>-6 | D<br>-5 | D1 | D 2 | D 3 | D 4 | D 5 | D 8 | W<br>2 | W 3 | <b>W</b> 4 | W 5 | 6 | | W<br>10 | W<br>1<br>2 | W<br>1<br>6 | | W<br>24 | | Every 6 | Withd |
| Visit Window | | n/a | n/a | n/a | n/a | n/ a | n/a | n/a | ±1 d | lay | | | | ±3 ( | days | | | | ±7 da | ays | | | | | ±14<br>days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 1<br>8 | 19 | 20 | 2 | 2 | 23 | 24 | 25-30 | 31+ | |
| Vector Copies<br>(Persistence) for<br>Research | | | X | | | | | X | X | | X | | X | X | | X | | | X | | X | | | | | | X |

Abbreviations: CARTOX = CAR T-Cell Treatment Toxicities; CMV = cytomegalovirus; CRP = C-reactive protein; CRS = cytokine release syndrome; CT = computerized tomography; ECG = electrocardiogram; ECHO = echocardiogram; ECOG = Eastern Cooperative Oncology Group; EDC = electronic data capture; FPCP = female patient of childbearing potential; GFR = glomerular filtration rate; MRI = magnetic resonance imaging; MUGA = multigated acquisition; n/a=not applicable; PCR = polymerase chain reaction; PFT = pulmonary function test; RCL = replication competent lentivirus; TSH = thyroid-stimulating hormone; VSV-G = vesicular stomatitis virus G protein

- Participants must have completed screening under Screening Protocol, ADP-0000-001, and confirmed as HLA-A\*02:01, HLA-A\*02:05, and/or HLA-A\*02:06 positive and have NY-ESO-1 and/or LAGE-1a positive tumor prior to conducting the procedures in this visit. <u>All</u> clinical assessments and procedures in this visit must be performed as indicated and recorded in source documents; however, only those assessments/procedures indicated with bold X<sub>EDC</sub> will be recorded in the EDC at this visit.
- 2. Refer to Section 5.2 (in protocol) for details on prophylaxis therapies, pre-medications, fludarabine dose adjustments according to renal function, and supportive treatments.
- 3. All samples will be collected and assessments performed prior to T-cell infusion, unless otherwise specified.
- 4. All clinical assessments required at the Screening visit must be performed within 28 days of leukapheresis, with the exception of lymphocyte subset (CD3/CD4/CD8), hematology, chemistry, coagulation and urinalysis which must be done within 7 days of leukapheresis. ECHO/MUGA, MRI/CT scan and laboratory assessments performed as standard of care prior to study consent will be acceptable as long as assessment is done within required time period before leukapheresis.
- 5. If a participant withdraws consent or completes the Interventional Phase 1, all procedures and assessments listed at this visit must be performed, unless done within the previous 30 days.
- 6. All clinical assessments and procedures must be performed as indicated; however, any clinical assessment or procedure can be performed if clinically indicated at any time
- Written participant informed consent must be obtained prior to performing any assessment or procedures, unless otherwise specified.
- 8. Participants must meet all eligibility prior to leukapheresis as specified in Section 4.2 (in protocol).

- 9. Participants must continue to meet all eligibility criteria (Section 4.2 (in protocol)) in addition to meeting those prior to lymphodepleting chemotherapy specified in Section 4.3 (in protocol)
- 10. Medical history will be recorded in the EDC at Screening and Baseline visits; however, any changes in medical history must be recorded in source documents throughout the conduct of the study.
- 11. Includes all prescription, over-the-counter medications, and herbal remedies. Any use of mutagenic agents or investigational agents must also be reported.
- 12. Includes temperature, blood pressure, pulse rate, respiratory rate, and oxygen saturation. Height will be collected at the Screening visit only.
- 13. Vital signs on day of T cell infusion should be taken pre-infusion, and at 5, 15 and 30 minutes, and 1, 1.5, 2, and 4 hours after the infusion has started
- 14. If a participant is found to have a tumor response or PD by imaging, a follow-up confirmation scan must be done no earlier than 4 weeks following the scan when response or PD first seen. A participant is not considered to have a response or PD until follow-up scan confirms the finding.
- 15. Includes FEV1, FVC, TLC, and DLCO parameters to determine eligibility as described in Exclusion criterion #23.
- <sup>16.</sup> FPCP must have a negative urine or serum pregnancy test.
- 17. Includes HIV, HBV, HCV, HTLV, EBV, and syphilis (spirochaete bacterium). Refer to Exclusion criterion #25 for details on required testing for eligibility. Testing for infectious disease markers is required only at Screening and does not need to be repeated at Baseline to satisfy eligibility criteria.
- 18. Only participants who are CMV IgG seropositive at Baseline will continue to be monitored for CMV viremia by CMV DNA PCR post Baseline.
- <sup>19.</sup> A free T4 test should be performed in participants who have an abnormal TSH function test (high or low).
- <sup>20.</sup> If CRS is suspected, cytokine and C-reactive protein levels should be measured approximately every other day until symptoms are improving or an alternative diagnosis is confirmed
- 21. Only to be done in participants ≥65 years of age to measure renal function.
- Adverse events should be reported as noted in Section 9 (in protocol)
- Persistence of gene modified cells in participants will be monitored at Months 3, 6, and 12 post-infusion, then every 6 months until 5 years post-infusion and annually from year 6-15 post infusion. If no gene modified cells are detected for 3 consecutive assessments post-infusion, and participant is ≥5 years post-infusion, then sample collection may stop.
- If RCL tests are negative at all time points during the first year, then samples will be collected annually and archived for up to 15 years post infusion or until assessments for persistence have ended. However, if VSV-G DNA copies are detected at any time point in the first year post-infusion, refer to the safety monitoring procedures in Section 10.1.2 (in protocol)
- <sup>25.</sup> If pharmacogenetic sample collection is not done at Baseline, it may be done at any other subsequent visit in the Interventional Phase 1. Collection of a pharmacogenetic sample is optional and all participants must provide consent for sample collection and analysis.
- <sup>26.</sup> Core needle biopsies for research are at Baseline, week 8, and at confirmation of PD, with the exception of participants for whom there is no safely accessible tumor tissue. 26a.) If a fresh biopsy was taken for NY-ESO-1and/or LAGE-1a confirmation screening in Screening Protocol, ADP-0000-001, and there is sufficient tumor sample left remaining, this sample may be used as the baseline sample. Otherwise, the Baseline biopsy may be collected anytime between two months and two weeks prior to the start of lymphodepleting chemotherapy, with preference closer to the time of infusion. 26b.) Exosome/cfDNA samples should match tumor biopsy time points.
- 27. Pre-infusion and Week 8 blood collection is for both Cytokine and Humoral anti-infused cell responses, and is collected in one 3 ml tube.
- <sup>28.</sup> Brain MRI (or CT Scan if MRI not feasible) should be obtained in all participants at the time of screening. Baseline brain MRI should be repeated if more than 4 months have elapsed prior to lymphodepletion.
- <sup>29.</sup> CARTOX-10 should be measured on the day of NY-ESO-1c259T cell infusion prior to receiving treatment and then at least through Day 8 according to the schedule of procedures. Participants with known brain metastases should be monitored at least twice per day for the first 5 days following NY-ESO-1c259T cell infusion. If a participant is found to have ES, the CARTOX-10 should be used at least twice per day until resolution or stable. It can also be used at later visits if indicated.

208749

## 14.2.2. Protocol Schedule of Events Interventional Phase II

## Table 4 Schedule of Procedures for Second T Cell Infusion (Interventional Phase 2)

| | | | Interve | ention | al Phas | se 2 | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline <sup>1</sup> | | Lymph<br>Chemo | | | T-cell in-<br>fusion <sup>3</sup> | Post | -T-ce | ll Inf | usion | | | | | | | | | | | Completion/<br>Withdrawal <sup>5</sup> |
| Day (D) / Week<br>(W) | -28 D <sup>4</sup> of<br>Chemo-<br>therapy | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D2 | D3 | D4 | D5 | D8 | W 2 | W 4 | W 8 | W<br>12 | W<br>16 | W 20 | W 24 | | Every 6 Mos<br>Thereafte r | |
| Visit Window | | n/a | n/a | n/a | n/a | n/a | ±1 d | ay | 1 | | 1 | ±3 da | ays | | ±7 d | ays | 1 | | ±14 days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 14 | 17 | 19 | 20 | 21 | 22 | 23-28 | 29+ | |
| | Clinical As | sessn | nents ai | nd Pro | ocedur | es <sup>6</sup> (refer t | o Sec | tion ' | 7.4 of | the p | rotoc | ol for | deta | ils) | | | • | | | | · |
| Informed<br>Consent <sup>7</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Inclusion/<br>Exclusion | X8 | | | | | | | | | | | | | | | | | | | | |
| Medical History <sup>9</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Physical Exam | X | | | | | X | | | | | X | X | | | | | | | | | |
| Prior/Concomitant Medications 10 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECOG | X | | | | | X | | | | | X | X | X | X | X | X | | X | X | X | X |
| Vital Signs /<br>Height/ Weight 11 | X | | | | | X <sup>12</sup> | X | X | X | X | X | X | | | | | | | | | X |
| ECG | X | | | | | X | | | X | | X | | | | | | | | | | |

| | | | Interve | mti an | al Dha | | | | | | | | | | | | | | | | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline <sup>1</sup> | | Lymph<br>Chemo | odep | leting | T-cell in-<br>fusion <sup>3</sup> | Post- | T-cel | l Infu | sion | | | | | | | | | | | Completion/<br>Withdrawal <sup>5</sup> |
| | -28 D <sup>4</sup> of<br>Chemo-<br>therapy | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D2 | D3 | D4 | D5 | D8 | W 2 | W 4 | W 8 | W 12 | 2W 16 | 6W 20 | W 24 | Every 3<br>Mos Until<br>Yr 2. | Every 6 Mos<br>Thereafter | |
| Visit Window | | n/a | n/a | n/a | n/a | n/a | ±1 da | ay | | <u> </u> | <u> </u> | ±3 d: | ays | | ±7 d | ays | | | ±14 days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 14 | 17 | 19 | 20 | 21 | 22 | 23-28 | 29+ | |
| ECHO/MUGA | X | | | | | | | | | | | | | | | | | | | | |
| CT / MRI <sup>13</sup> | X | | | | | | | | | | | | | X | | X | | X | X | X | X |
| Brain MRI | X | | See foo | tnote | 27 | • | | | | | | | | | 1 | | 1 | | | • | • |
| Chest X-ray | X | | | | | | | | | | | | | | | | | | | | |
| PFTs <sup>14</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Lymphocyte<br>subset<br>(CD3/CD4/CD8) | Х | | | | | | | | | | | | | | | | | | | | |
| Hematology | X <b>4</b> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Chemistry | X <b>4</b> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | X | X |
| Coagulation Tests | X <b>4</b> | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test <sup>15</sup> | X | X | | | | X | | | | | | | X | X | X | X | X | X | X | X | X |
| Urinalysis | X <b>4</b> | | | | | | | | | | | | | | | | | | | | |
| Infectious disease markers 16 | X | | | | | | | | | | | | | | | | | | | | |

| | | | Interv | ention | al Phas | se 2 | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline <sup>1</sup> | | Lympl | | | T-cell in- | Dogt | T col | l Infu | a <b>i</b> an | | | | | | | | | | | Completion/ |
| | Dascinic | | Chemo | othera | ipy <sup>2</sup> | fusion <sup>3</sup> | rost- | · 1 -cei | 1 1111u | SIOH | | | | | | | | | | | Withdrawal <sup>5</sup> |
| Day (D) / Week<br>(W) | -28 D <sup>4</sup> of<br>Chemo-<br>therapy | D<br>-8 | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D2 | D3 | D4 | D5 | D8 | W 2 | W 4 | W 8 | W 1 | 2 W 1 | 6 W 2 | 20 W 24 | Every 3 Mos<br>Until Yr 2. | Every 6<br>Mos<br>Thereafter | |
| Visit Window | | n/a | n/a | n/a | n/a | n/a | ±1 da | ay | 1 | 1 | 1 | ±3 d | lays | | ±7 d | ays | | | ±14 days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 14 | 17 | 19 | 20 | 21 | 22 | 23-28 | 29+ | |
| Fludarabine | | X | X | X | X | | | | | | | | | | | | | | | | |
| Cyclophos-<br>phamide | | | X | X | X | | | | | | | | | | | | | | | | |
| NY-ESO-1 <sup>c259</sup> T | | | | | | X | | | | | | | | | | | | | | | |
| | Correlative | Stud | ies and | Resea | rch As | sessments | (refer | to Se | ction | 7.5 of | the P | rotoco | ol for | detail | ls) | | | | 1 | • | • |
| Tumor biopsy <sup>25</sup> | X <sup>25</sup> a | | | | | | | | | | | | | X | | | | | | | X |
| Liquid biopsy <sup>25</sup> | X | | | | | X | | | | | X | | X | X | | X | | | | | X |
| Cell phenotype<br>and Functional | | | | | | X | | | X | | X | X | X | X | X | | | | $X^{28}$ | X <sup>28</sup> | X |
| Assays,<br>Cytokine | | | 1 | | | <sub>X</sub> 26 | X | X | X | X | X | X | X | 26 | v | - | - | | $X^{28}$ | X <sup>28</sup> | X |
| Analyses 19 | | | | | | X20 | Λ | Λ | Λ | Λ | Λ | Λ | Λ | X26 | Λ | | | | Λ | Λ | Λ |
| & Humoral Anti-<br>Infused Cell | | | | | | | | | | | | | | | | | | | | | |
| Responses | | | | | | | | | | | | | | | | | | | | | |

208749

| | Baseline <sup>1</sup> | | Interve<br>Lymph<br>Chemo | odepl | eting | T-cell in- | | T-cel | l Infus | sion | | | | | | | | | | | Completion/<br>Withdra<br>wal <sup>5</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (D) / Week<br>(W) | -28 D <sup>4</sup> of<br>Chemo-<br>therapy | | <b>D</b><br>-7 | D<br>-6 | D<br>-5 | D1 | D2 | D3 | D4 | D5 | D8 | W 2 | W 4 | W 8 | W 12 | W 16 | W 20 | W 24 | Every 3 Mos<br>Until Yr 2. | Every 6 Mos<br>Thereafter | |
| Visit Window | | n/a | n/a | n/a | n/a | n/a | ±1 da | ıy | ı | | 1 | ±3 da | ys | | ı | ±7 da | ys | 1 | ±14 days | ±3 mos | n/a |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 14 | 17 | 19 | 20 | 21 | 22 | 23-28 | 29+ | |
| Vector Copies<br>(Persistence) for<br>Research | X <sup>1</sup> | | | | | X | X | | X | | X | X | X | X | X | X | | | | | X |

Abbreviations: CMV = cytomegalovirus; CRP = C-reactive protein; CRS = cytokine release syndrome; CT = computed tomography; ECG = electrocardiogram; ECHO = echocardiogram; ECOG = Eastern Cooperative Oncology Group; FPCP = female patient of childbearing potential; MRI = magnetic resonance imaging; n/a=not applicable; PCR = polymerase chain reaction; PFT = pulmonary function test; RCL = replication competent lentivirus; TSH = thyroid-stimulating hormone; VSV-G = vesicular stomatitis virus G protein

- 1. Participants must have been considered eligible for a second infusion (refer to Section 4.4 (in protocol)) before initiating any screening procedures or assessments for Interventional Phase 2.
- Refer to Section 5.2 (in protocol) for details on prophylaxis therapies, pre-medications, fludarabine dose adjustments according to renal function, and supportive treatments.
- 3. All samples will be collected and assessments performed prior to T-cell infusion, unless otherwise specified.
- 4. Clinical procedures or assessments do not need to be repeated at this Baseline visit if they were be performed within 28 days of planned leukapheresis, with the exception of lymphocyte subset (CD3/CD4/CD8), hematology, chemistry, coagulation and urinalysis which must be done within 7 days of leukapheresis.
- If a participant withdraws consent or completes the Interventional Phase 2, all procedures and assessments listed at this visit must be performed, unless done within the previous 30 days.
- 6. All clinical assessments and procedures must be performed as indicated; however, any clinical assessment or procedure can be performed if clinically indicated at any time.
- An additional written participant informed consent for a second infusion must be obtained prior to performing any Baseline assessments or procedures, unless otherwise specified.

- Participants must continue to meet all eligibility criteria (Section 4.2 and Section 4.3 (in protocol)) in addition to meeting those prior to second infusion specified in Section 4.4 (in protocol)).
- 9. Any new or changes in medical history will be recorded in the EDC at Baseline visit; however, any additional changes in medical history must be recorded in source documents throughout the conduct of the study.
- 10. Includes all prescription, over-the-counter medications, and herbal remedies. Any use of mutagenic agents or investigational agents must also be reported.
- 11. Includes temperature, blood pressure, pulse rate, respiratory rate, and oxygen saturation. Height will be collected at the Screening visit only.
- 12. Vital signs on day of T cell infusion should be taken pre-infusion, and at 15 and 30 minutes, and 1, 1.5, 2, and 4 hours after the infusion has started.
- 13. If a participant is found to have a tumor response or PD by imaging, a follow-up confirmation scan must be done no earlier than 4 weeks following the scan when response or PD first seen. A participant is not considered to have a response or PD until follow-up scan confirms the finding.
- 14. Includes FEV1, FVC, TLC, and DLCO parameters to determine eligibility as described in Exclusion criterion #23.
- 15. FPCP must have a negative urine or serum pregnancy test.
- 16. Includes HIV, HBV, HCV, HTLV, EBV, and syphilis (spirochaete bacterium). Refer to Exclusion criterion #25 for details on required testing for eligibility.
- 17. Only participants who are CMV IgG seropositive at baseline will continue to be monitored for CMV viremia by CMV DNA PCR post baseline.
- <sup>18.</sup> A free T4 test should be performed in participants who have an abnormal TSH function test (high or low).
- 19. If CRS is suspected, cytokine and C-reactive protein levels should be measured approximately every other day until symptoms are improving or an alternative diagnosis is confirmed.
- Only to be done in participants  $\geq$ 65 years of age to measure renal function.
- <sup>21</sup>. Adverse events should be reported as noted in Section 9 (in protocol).
- Persistence of gene modified cells in participants will be monitored at Months 3, 6, and 12 post-infusion, then every 6 months until 5 years post-infusion and annually from year 6-15 post infusion. If no gene modified cells are detected for 3 consecutive assessments post-infusion, and participant is >5 years post-infusion, then sample collection may stop.
- <sup>23</sup> If RCL tests are negative at all time points during the first year, then samples will be collected annually and archived for up to 15 years post or until assessments for persistence have ended However, if VSV-G DNA copies are detected at any time point in the first year post-infusion, refer to the safety monitoring procedures in Section 10.1.2 (in protocol).
- <sup>24.</sup> CARTOX-10 should be measured on the day of NY-ESO-1c259T cell infusion prior to receiving treatment and then at least through Day 8 according to the schedule of procedures. Participants with known brain metastases should be monitored at least twice per day for the first 5 days following NY-ESO-1c259T cell infusion. If a participant is found to have ES, the CARTOX-10 should be used at least twice per day until resolution or stable. It can also be used at later visits if indicated.
- <sup>25.</sup> Core needle biopsies are at baseline, week 8, and at confirmation of PD, with the exception of participants for whom there is no safely accessible tumor tissue. 24a.) If a fresh biopsy was taken to confirm continued expression of NY-ESO-1 and/or LAGE-1a at the time of PD after the first T cell infusion and there is sufficient tumor sample left remaining, this sample may be used as the baseline sample. Otherwise, the baseline biopsy may be collected anytime between two months and two weeks prior to the start of lymphodepleting chemotherapy, with preference closer to the time of infusion. 24b.) Exosome/cfDNA samples should match tumor biopsy time points.
- <sup>26</sup>. Pre-infusion and Week 8 blood collection is for both Cytokine and Humoral anti-infused cell responses, and is collected in one 3 ml tube.
- 27. Brain MRI will be performed at baseline for all participants and as clinically indicated thereafter (see Section 8.9.2 (in protocol)).

208749

## 14.2.3. Protocol Defined Schedule of Events Long Term Follow-up

## Table 5 Schedule of Procedures – Long Term Follow- up

| Time post-infusion | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Year 1 | | | Year 2 | 2 | Year | 3 | Year 4 | 4 | Year | 5 | Years 6-15 |
| Months | 3 | 6 | 12 | 18 | 24 | 30 | 36 | 42 | 48 | 54 | 60 | Annually |
| Visit window | ± 2 we | eks | ± 3 mo | nth | | | | L | <u> </u> | | <b>I</b> | ± 6 months |
| Safety Assessments | • | | <b>I</b> | | | | | | | | | • |
| Medical History and Physical Exam <sup>1</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Mutagenic agents, other investigational agents or anti-cancer therapies | | X | X | X | X | X | X | X | X | X | X | X |
| Delayed adverse Events and Serious Adverse Events <sup>2</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test for WOCBP <sup>3</sup> | <==== | | | | X | 3 | | | | ===> | • | • |
| Hematology | | X | X | | X | | X | | X | | X | X <sup>4</sup> |
| Serum chemistry | | X | X | | X | | X | | X | | X | X <sup>4</sup> |
| Allogeneic SCT | X | X | X | X | X | | | | | | | |
| Laboratory Assessments | | | | | | | | | | | | |
| VSV-G DNA (RCL) for safety | X | X | X | | X | | X | | X | | X | X <sup>4</sup> |
| Transgene Copies (Persistence) for safety | X | X | X | X | X | X | X | X | X | X | X | X |
| Other Assessments | 1 | 1 | 1 | | 1 | 1 | ı | | ı | 1 | 1 | L |
| Survival Status | X | X | X | X | X | X | X | X | X | X | X | X |

Abbreviations: RCL=replication competent lentivirus; SCT=stem cell transplant; VSV-G=vesicular stomatitis virus G protein

<sup>1.</sup> New medical history/medications/chemotherapies.

<sup>2.</sup> Delayed adverse Event and Serious Adverse Event collection is limited to:

<sup>☐</sup> New malignancies

208749

New incidence or exacerbation of a pre-existing neurologic disorder
 New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder
 New incidence of immune-related hematologic disorder
 Serious infections (including opportunistic)
 Unanticipated illness and/or hospitalization deemed related to gene modified cell therapy
 For women of child bearing potential (WOCBP), pregnancy testing should be conducted during contraception period only as defined in Section 5.1 (in protocol). When pregnancy testing is performed at visits where hematology sample is collected, blood pregnancy testing will be done. At visits where hematology sample is not collected, urine pregnancy test is acceptable unless serum testing is required by local regulation or IRB/IEC.

4. In year 6-15, these assessments are performed for as long as persistence is analyzed. If persistence samples are discontinued (Section 10.3 (in protocol)) then laboratory assessments are discontinued

208749

## 14.3. Appendix 3: Assessment Windows

Assessment windows will not be used.

# 14.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 14.4.1. Study Phases

#### 14.4.1.1. Study Phases for Concomitant Medications

| Study Phase | Definition |
|---|---|
| Prior | End date of medication is not missing and is before the start date of lymphodepletion |
| | OR lymphodepletion start date is missing |
| Concomitant | Medication is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Datafor handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is missing.

#### 14.4.1.2. Study Phases for Anti-Cancer Therapy/Surgery

| Study Phase | Definition |
|---|---|
| Prior | Start date is prior to first day of leukapheresis or leukapheresis start date is missing |
| Bridging | Start date is on or after the day of apheresis to the day before initiation of lymphodepletion chemotherapy |
| On-Study | Start date is on or after the first day of lymphodepletion chemotherapy |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for anti-cancer therapy

## 14.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after first lymphodepletion chemotherapy start date.<br/>(Lymphodepletion Start Date ≤ AE Start Date) until end of study, include AEs onset on or after the second lymphodepletion for participants who receive a second T-cell infusion.</li> </ul> |
| | <ul> <li>Treatment emergence for second infusion will be defined as: If AE onset date is<br/>on or after second lymphodepletion chemotherapy start date.<br/>(Lymphodepletion Start Date ≤ AE Start Date) until end of study.</li> </ul> |
| | If AE onset date is missing and AE end date is before the lymphodepletion start date, then the AE will not be classified as Treatment-Emergent. If AE onset date is missing and AE end date is either missing or on or after lymphodepletion start date, then the AE will be classified as treatment-emergent A E OF A COLOR OF A CO |
| | <ul> <li>Missing AE Start Date will be imputed following rules in Section 14.7.2.1 for<br/>determining Treatment Emergent AEs.</li> </ul> |

208749

## 14.5. Appendix 5: Data Display Standards & Handling Conventions

## 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound | : arprod\GSK3377794\mid208749 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1].</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for SAC upon request. | |

## 14.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All participant level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

| Unscheduled Visits | |
|---|---|
| | <ul> <li>Unscheduled visits will not be included in summary tables and/or figures, except in cases where<br/>worse-case post-baseline is calculation.</li> </ul> |
| All unscheduled v | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

208749

### 14.6. Appendix 6: Derived and Transformed Data

#### 14.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- For character variables, if multiple assessments on different days are reported for the same scheduled assessment, then the worst case assessment for that scheduled assessment will be analyzed
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from T cell infusion date:
  - Ref Date = Missing → Study Day = Missing
  - o Ref Date < T cell infusion Date → Study Day = Ref Date T cell infusion Date
  - o Ref Data ≥ T cell infusion Date → Study Day = Ref Date T cell infusion Date + 1

Second study day (Study Day 2) will be calculated for participants with second T-cell infusion as below

- Ref Date = Missing → Study Day = Missing
- Ref Date < Second T cell infusion Date → Study Day = Ref Date Second T cell infusion Date</p>
- Ref Data ≥Second T cell infusion Date → Study Day = Ref Date Second T cell infusion Date
   + 1

#### Change from Baseline

- Change from Baseline = Post-Baseline Visit Value Baseline
- % Change from Baseline= 100 x (Post-Baseline Visit Value Baseline) / Baseline
- Maximum Increase/Decrease from Baseline = maximum (Increase/Decrease from Baseline)
- If either the Baseline or Post-Baseline Visit Value is missing, Change from Baseline and % Change from Baseline is set to missing

#### **Date of Response**

For post-baseline disease assessments, the date of response (PR,CR) is assigned to the latest date
of disease assessments; for other response categories (SD, NE, PD), the date of response is
assigned to the earliest date of disease assessments.

### **Date of New On-study Anti-Cancer Therapy**

- Derived as the earliest date of new on-study anti-cancer therapy, radiotherapy (where applicable) or cancer-related surgical procedure (where applicable)
- Missing or partial dates will be imputed for derivation of new anti-cancer therapy following rules specified in Section 14.7.2.1.

208749

#### 14.6.2. Study Population

#### Age

 For participants with a T-cell infusion date, age is derived using T-cell infusion date as the reference date. For ITT participants without a T-cell Infusion date, date of eligibility for apheresis is used as the reference date.

#### **BMI**

(Weight in kg) / (Height in meters)<sup>2</sup>

#### **Time from Screening to Initial Diagnosis**

- Calculated as the number of months from the Date of Initial Diagnosis:
  - Informed Consent Date = Missing → Elapse Time = Missing
  - Date of Initial Diagnosis = Completely/partially Missing → Elapse Time = Missing
- Otherwise → Elapse Time = (Informed Consent Date Date of Initial Diagnosis + 1)/30.4375

## 14.6.3. Efficacy

Refer to Section 7 for endpoint derivation information.

#### **Overall Survival**

#### **Date of Last Contact**

- Last date in all SDTM domains
- If patient died, the last contact date should be death date.
- Dates after date of death will be excluded. Future dates will be excluded.
- SDTM domain SE and SUPPBE will be excluded and SDTM variables DM.BRTHDTC, MH.MHSTDTC, SV.SVENDTC, SV.SVSTDTC, DM.RFPENDTC, \_ALL\_.ANALDTC, DV.DVDTC, DV.DVSTDTC, and RS.RSDTC where RSEVAL='INDEPENDENT ASSESSOR' will be excluded
- Partial and missing dates will not be imputed for the purpose of deriving date of last contact

208749

#### 14.6.4. Safety

#### **Adverse Events**

#### **AE'S of Special Interest**

- Cytokine Release Syndrome
- Pneumonitis
- Graft vs Host Disease
- Haematopoietic cytopenias (including pancytopenia and aplastic anaemia)
- Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS)
- Guillain-Barre Syndrome

#### **Duration of AE**

- Calculated as the number of days from AE Start Date to AE Stop Date:
  - $\circ$  AE Start Date = Missing  $\rightarrow$  Elapse Time = Missing
  - AE Stop Date = Missing → Elapse Time = Missing

Otherwise → Elapsed Time = AE Stop Date – AE Start Date + 1 Imputed dates will not be used to calculated AE duration

## **Corrected Calcium for Albumin**

- Corrected Calcium [mg/dL] = Total Calcium [mg/dL] + 0.8 \* (4.0 serum albumin [g/dL])
- Corrected Calcium [mmol/L] =
   Total Calcium [mmol/L] / .2495 + 0.8 \* .2495 \* (4.0 serum albumin [g/L]/10)

## 14.7. Appendix 7: Reporting Standards for Missing Data

## 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as when<br/>he/she has PD or has died prior to PD, or 2 years after the NY-ESO T-cell infusion,<br/>whichever is shorter for participants that receive one T-cell infusion. For participants<br/>that receive a second T-cell infusion, study completion is defined as when he/she has<br/>PD or has died prior to PD, or 6 months after the second T-cell infusion, whichever is<br/>shorter.</li> </ul> |
| | Withdrawn participants were not replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

## 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing<br/>displays. Unless all data for a specific visit are missing in which case the data<br/>is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays. However,<br/>where necessary, display macros may impute dates as temporary variables for<br/>sorting data in listings only. In addition, partial dates may be imputed for 'slotting'<br/>data to study phases (see Section 14.4.1) or for specific analysis purposes as<br/>outlined below.</li> </ul> |
| | <ul> <li>Imputed partial dates will not be used to derive study day, duration (e.g., duration of adverse events), or elapsed time variables unless otherwise specified. In addition, imputed dates are not used for deriving the last contact date in overall survival analysis dataset.</li> </ul> |
| | <ul> <li>Imputed partial dates for anti-cancer therapy, surgery, and radiotherapy will be<br/>used for plotting therapies in Figure 3.010, only if the day is missing.</li> </ul> |
| Adverse Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>This includes identifying an AESI as first or last occurrence.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | Missing start day | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = 1st of month.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If month and year of start date = month and year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = 1st of month.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month Missing stop day | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = January 1.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If year of start date = year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = January 1.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = January 1.</li> </ul> </li> <li>Last day of the month will be used.</li> </ul> |
| | Missing stop day and month | No Imputation |
| | Completely missing start/end date | No imputation. |
| Concomitant<br>Medications | The state of the | |
| | Missing start day | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not receive lymphodepletion), then set start date = 1st of month.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If month and year of start date = month and year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = 1st of month.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | If lymphodepletion start date is missing (i.e. participant did not receive lymphodepletion), then set start date = January 1. |

| | eporting Detail | Else if lymphodepletion start date is not missing: |
|---|---|---|
| M<br>a<br>C | Missing end day Missing end day and month Completely missing start/end date | <ul> <li>If year of start date = year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = January 1.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = January 1.</li> <li>A '28/29/30/31' will be used for the day (dependent on the month and year)</li> <li>A '31' will be used for the day and 'Dec' will be used for the month.</li> <li>No imputation</li> </ul> |
| Anti-Cancer Therapy and Radiotherapy • | Completely missing applied. If partial start date of the start da | ng start or end dates will remain missing, with no imputation e contains a year only set to January 1st. e contains a month and year set to the 1st of the month. partial end dates will be performed. |
| Surgical Procedures • | If partial date contains a year only set to January 1st. | |
| New On-study Anti-Cancer Therapy/ Radiotherapy/ Surgical Procedures for Efficacy Evaluation | surgical procedur define event and duration of respon be imputed when following rules will on anti-cancer the Completely missis Partial start dates If both month If only day is If the month day; If the month assessm date of control the day; If both control Otherwise | onth of partial date is the same as the month of T-cell infusion, on of (T-cell infusion + 1, last day of the month) will be used for the onth of partial date is the same as the month of last disease ment and the last disease assessment is PD, minimum of (last disease assessment + 1, last day of the month) will be used for |

### 14.8. Appendix 8: Values of Potential Clinical Importance

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 4.03) will be used to assign grades for laboratory parameters including clinical chemistry, hematology, liver function tests, thyroid function tests, pancreatic enzyme tests, QTc (Bazett's or Fridericia's) values, and vital signs (heart rate, blood pressure, temperature).

## 14.8.1. Laboratory Values

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03) will be used to assign grades to the relevant laboratory parameters. NCI-CTCAE v4.03 can be found at http://ctep.cancer.gov/reporting/ctc.html.

For laboratory data which are not listed in the NCI CTCAE v4.03, a summary of values outside the normal range will be provided.

For lab test values that can be graded, values of grade 1 or above are defined as values of potential clinical concern. For lab test values that cannot be graded, values out of the normal range are defined as values of potential clinical concern. Abnormal, clinically significant Urinalysis labs will be also be considered PCI values.

#### 14.8.2. ECG Parameters

To identify QTc (Bazett's or Fridericia's) values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign grades (see adverse event 'Electrocardiogram QT corrected interval prolonged'). The CRF collects either QTcB or QTcF. Note that there is a slight inconsistency between CTCAE v4.03 and ICH E14 (Absolute QTc interval prolongation). It was decided to align with CTCAE for the oncology standard categories.

The following criteria will be used to flag electrocardiogram (ECG) values that are values of potential clinical importance:

208749

| PCI Flag | Potential Clinical Importance (PCI) Range |
|---|---|
| High (H) | Grade 2 or Higher (QTc>480)<br>or<br>QTc increase from baseline of >30msec |

## 14.8.3. Vital Signs

To identify heart rate values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Sinus bradycardia', 'Sinus tachycardia', 'Supraventricular tachycardia', and 'Ventricular tachycardia'.

The following criteria will be used to flag vital sign values that are values of potential clinical importance:

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Decrease from baseline<br>Heart Rate | Decrease to <60 | bpm |
| Increase from baseline<br>Heart Rate | Increase to >100 | bpm |

To identify blood pressure values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypertension'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|-------------------------|-------------------------------------------|------|
| Increase from baseline | ≥120 to <140 (Grade 1) | mmHg |
| Systolic Blood Pressure | ≥140 to <160 (Grade 2) | |
| | ≥160 (Grade 3) | |
| Increase from baseline | ≥80 to <90 (Grade 1) | mmHg |
| Diastolic Blood | ≥90 to <100 (Grade 2) | |
| Pressure | ≥100 (Grade 3) | |

To identify temperature values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypothermia' and 'Fever'.

## 208749 | Statistical Analysis Plan RAP 02 Oct 2020 | TMF-2069301 | 1.0

#### CONFIDENTIAL

208749

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|------------------------|-------------------------------------------|---------|
| Increase from baseline | Increase to ≥38 | Degrees |
| temperature | | C |
| Decrease from baseline | Decrease to ≤35 | Degrees |
| Diastolic Blood | | C |
| Pressure | | |

To identify oxygen saturation values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with "Hypoxia"

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|-----------------------|-------------------------------------------|------|
| Decrease for baseline | Decrease to <88 | % |
| oxygen saturation | | |

208749

## 14.9. Appendix 9: Abbreviations & Trade Marks

## 14.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CRS | Cytokine Release Syndrome |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOR | Duration of Response |
| DP | Decimal Places |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| GvHD | Graft versus Host Disease |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LVEF | Left Ventricular Ejection Fraction |
| MedDRA | Medical Dictionary for Regulatory Affairs |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| PCI | Potential Clinical Importance |
| PFS | Progression Free Survival |
| PP | Per Protocol |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |

208749

| Abbreviation | Description |
|--------------|------------------------------|
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TTR | Time to Response |
| WHO | World Health Organization |

## 14.9.2. Trademarks

| Traden | narks of the GlaxoSmithKline<br>Group of Companies |
|--------|----------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
208749

#### 14.10. Appendix 10: List of Data Displays

#### 14.10.1. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays. Shells are subject to some minor formatting modifications post RAP approval.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Biomarker | BIO_Fn | BIO_Tn | BIO_Ln |

#### NOTES:

#### 14.10.2. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|----------------|----------------|
| Study Population | 1.010 to 1.320 | NA |
| Efficacy | 2.010 to 2.080 | 2.010 to 2.050 |
| Safety | 3.010 to 3.670 | 3.010 to 3.040 |
| Pharmacodynamic and / or Biomarker | 6.010 to 6.020 | 6.010 to 6.290 |
| Section | List | ings |
| ICH Listings | 10 to 580 | |
| Other Listings | 590 t | o 680 |

#### 14.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------|
| SAC | Statistical Analysis Complete |

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 208749

# 14.10.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subject | Subject Disposition | | | | |
| 1.010. | ITT | POP_T2 | Summary of Subject Status- Interventional Phase 1 (ITT Population) | ICH E3, FDAAA, EudraCT | SAC |
| 1.020. | mITT | POP_T2 | Summary of Subject Status- Interventional Phase 1 (mITT Population) | ICH E3, FDAAA, EudraCT | SAC |
| 1.030. | ITT | POP_T3 | Summary of Subject Status- End of Study | ICH E3, FDAAA, EudraCT | SAC |
| 1.040. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements Add a footnote that we only have data from about 40 subjects and x subjects were screened under Adaptimmune and why | SAC |
| 1.050. | ITT | NS1 | Summary of Number of Subject by Country and Site ID | EudraCT/Clinical Operations Include Site Name | SAC |
| 1.060. | ITT | Non-Standard | Summary of Apheresis, Lymphodepletion, and T cell Infusion | Use POP_T1 | SAC |
| Protoco | ol Deviation | | | | |
| 1.070. | ITT | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.080. | ITT | SP1A | Summary of Study Populations | IDSL<br>ITT, mITT, Second T-cell Infusion | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.090. | ITT | DM1 | Summary of Demographic Characteristics (ITT Population) | ICH E3, FDAAA, EudraCT Report baseline height, weight, and BMI, Report Race not Race Detail | SAC |
| 1.100. | mlTT | DM1 | Summary of Demographic Characteristics (mITT Population) | ICH E3, FDAAA, EudraCT Report screening height, weight, and BMI Report Race not Race Detail | SAC |
| 1.110. | ITT | DM11 | Summary of Age Ranges | EudraCT | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.120. | ITT | MH1 | Summary of Medical Conditions (ITT Population) | ICH E3 | SAC |
| 1.130. | mITT | MH1 | Summary of Medical Conditions (mITT Population) | ICH E3 | SAC |
| 1.140. | mITT | CM8 | Summary of Concomitant Medications | ICH E3<br>Use GSKDRUG | SAC |
| Exposu | re and Treatm | ent Compliance | | | |
| 1.150. | mlTT | OEX1 | Summary of Total Transduced T cells (First Infusion) | Report total number of transduced T cells in 10^9 cells and categorize it into < 1, >=1 to <=8, and >8 | SAC |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Disease | Disease Characteristics | | | | |
| 1.160. | ITT | DC1 | Summary of Disease Characteristics at Initial Diagnosis (ITT Population) | ICH E3 Time since initial diagnosis in months Stage of lung cancer at initial diagnosis Histology | SAC |
| 1.170. | mITT | DC1 | Summary of Disease Characteristics at Initial Diagnosis (mITT Population) | ICH E3 Time since initial diagnosis in months Stage of lung cancer at initial diagnosis Histology | SAC |
| 1.180. | ITT | DC2 | Summary of Disease Characteristics at Screening (ITT Population) | ICH E3 Disease stage at enrolment Tumor type Anatomical location NY-ESO-1 status HLA status Number of prior radiotherapy regimens (prior to leukapheresis – see study phase) Number of prior systemic therapy regimens (prior to leukapheresis- see study phase) | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.190. | mITT | DC2 | Summary of Disease Characteristics at Screening (mITT Population) | ICH E3 Disease stage at enrolment Tumor type Anatomical location NY-ESO-1 status HLA status Number of prior radiotherapy regimens (prior to leukapheresis – see study phase) Number of prior systemic therapy regimens (prior to leukapheresis- see study phase) | SAC |
| 1.200. | mITT | LA1 | Summary of Disease Burden at Baseline-First Infusion | ICH E3 Include target and non target lesions | SAC |
| Anti-Ca | ncer Therapy | | | | |
| 1.210. | ITT | AC1 | Summary of Prior Anti-Cancer Therapy (ITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |
| 1.220. | mITT | AC1 | Summary of Prior Anti-Cancer Therapy (mITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |
| 1.230. | mITT | FAC1 | Summary of On-Study Anti-Cancer Therapy | IDSL Add time from T-cell infusion to first post-treatment anti-cancer therapy, min, 25th Q, median, 75th Q, max | SAC |
| 1.240. | ITT | CM1 | Summary of Prior Dictionary Coded Anti-Cancer Therapy (ITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |

| Study Population Tables | | | | |
|---|---|---|---|---|
| Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| mITT | CM1 | Summary of Prior Dictionary Coded Anti-Cancer Therapy (mITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |
| mITT | CM1 | Summary of On-Study Dictionary Coded Anti-Cancer Therapy | IDSL | SAC |
| ITT | AC3 | Summary of Number of Anti-Cancer Therapy Regimens Prior to Leukapheresis (ITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |
| mITT | AC3 | Summary of Number of Anti-Cancer Therapy Regimens Prior to Leukapheresis (mITT Population) | IDSL Therapy before leukapheresis-see study phase | SAC |
| I/Medical Proc | edures | | | |
| ITT | OSP1 | Summary of Prior Cancer-Related Surgical Procedures (ITT Population) | IDSL Summarize like below; Any surgery Surgery Intent Curative, diagnostic, palliative, other Site of surgery Lobectomy, etc, other. | SAC |
| | Population mITT mITT ITT mITT | Population IDSL / Example Shell | Population IDSL / Example Shell Title | Population IDSL / Example Shell Title Programming Notes |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.300. | mITT | OSP1 | Summary of Prior Cancer-Related Surgical Procedures (mITT Population) | IDSL Summarize like below; Any surgery Surgery Intent Curative,diagnostic,palliative, other Site of surgery Lobectomy,etc,other. Surgery before leukapheresis | SAC |
| 1.310. | mITT | OSP1 | Summary of On-Study Cancer-Related Surgical Procedures | IDSL Summarize like below; Any surgery Surgery Intent Curative, diagnostic, palliative, other Site of surgery Lobectomy, etc, other. | SAC |
| Substa | Substance Use | | | | |
| 1.320. | mITT | SU1 | Summary of Substance Use | IDSL Cigarette use: smoking history, years smoked, packs per day | SAC |

208749

## 14.10.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respor | se Rate | | | | |
| 2.010. | mITT | RE1a | Summary of Investigator-Assessed Best Response with Confirmation (RECIST 1.1 Criteria) (mITT Population) – First Infusion | First infusion Do not keep: Best Response-Non-CR/Non-PD, Response Rate-p-value, or the last three sections (response rate, odds ratio, test for homogeneity). | SAC |
| | | | | Include footnote identify subject that does not have target lesion at baseline | |
| 2.020. | ITT | RE1a | Summary of Investigator-Assessed Best Response with Confirmation (RECIST 1.1 Criteria) (ITT Population)– First Infusion | First infusion Do not keep: Best Response-Non-CR/Non-PD, Response Rate-p-value, or the last three sections (response rate, odds ratio, test for homogeneity). | SAC |
| | | | | Include footnote identify subject that does not have target lesion at baseline | |
| 2.030. | mITT | RE1c | Summary of Investigator-Assessed Disease Control Rate with Confirmation (RECIST 1.1 Criteria) (mITT Population)– First Infusion | First infusion Do not keep any optional sections: Non-CR/Non-PD, P-value, or last 3 sections | SAC |
| | | | | Include footnote identify subject that does not have target lesion at baseline | |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.040. | ITT | RE1c | Summary of Investigator-Assessed Disease Control Rate with Confirmation (RECIST 1.1 Criteria) (ITT Population)– First Infusion | First infusion Do not keep any optional sections: Non-CR/Non-PD, P-value, or last 3 sections Include footnote identify subject that does not have target lesion at baseline | SAC |
| Time-to | -<br>-Event Endpoi | ints | | does not have target resion at basenine | |
| 2.060. | mITT | TTE1 | Summary of Progression-Free Survival by Investigator (RECIST 1.1 Criteria)– First Infusion | Only present Endpoint(Event) and Censored, do not include follow-up ended/ongoing. Remove hazard ratio, and log rank sections. Include footnote identify subject that does not have target lesion at baseline | SAC |
| 2.080. | mITT | TTE1 | Summary of Overall Survival | Only present Endpoint(Event) and Censored, do not include follow-up ended/ongoing. Remove Event summary, hazard ratio, and log rank sections. | SAC |

208749

## 14.10.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respor | se Rate | | | | |
| 2.010. | mITT | RE8b | Investigator-Assessed Maximum Percent Reduction from Baseline in Tumor Measurement (RECIST 1.1 Criteria)– First Infusion | Label with subject ID Include footnote identify subject that does not have target lesion at baseline | SAC |
| 2.020. | mITT | Non-Standard | Spider Plot of Percent Change from Baseline in Target Lesion<br>Diameter– First Infusion | Label with subject ID Use EFF_F1 Include footnote identify subject that does not have target lesion at baseline | SAC |
| Time-to | -Event Endpoi | ints | | | |
| 2.030. | mITT | TTE10 | Graph of Kaplan Meier Survival Curves of Progression-Free Survival with 95% Confidence Bands (RECIST 1.1 Criteria) – First Infusion | Include footnote identify subject that does not have target lesion at baseline | SAC |
| 2.050. | mITT | TTE10 | Graph of Kaplan Meier Survival Curves of Overall Survival with 95% Confidence Bands | | SAC |

208749

## 14.10.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.010 | ITT | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 Do not use combined PT Terms | SAC |
| 3.020 | mITT | AE1 | Summary of All Treatment Emergent Adverse Events by<br>System Organ Class and Preferred Term | ICH E3 Do not use combined PT Terms | SAC |
| 3.030 | ITT | AE1 | Summary of Adverse Events Grouped by Similarity of Preferred Terms | Only include combined PT term AEs -Remove "Any Event" row -SOC from AE1 should be Combined Term -PT term from AE1 should Preferred Term Label column "Synoymn/Preferred Term" If combined AE does not appear, include a 0 count. | SAC |
| 3.040 | ITT | OAE07 | Summary of All Adverse Events by Maximum Grade | Use Combined PT list FOR ALL COMBINED PT TABLES FOOTNOTE=Adverse Events are combined as showed in Table 3.40" COLUMN LABEL=Adverse Events All tables by maximum grade should only include Grade 3+4+5 column as in OAE01, not Grade 3+4 columns | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.050 | mITT | OAE07 | Summary of All Treatment Emergent Adverse Events by Maximum Grade | Use Combined PT list | SAC |
| 3.060 | mITT | OAE07 | Summary of All Study-Treatment Related Adverse Events by Maximum Grade | ICH E3 Use Combined PT list Treatment related including all lymphodepletion regimens and T-cell Infusion | SAC |
| 3.070 | mITT | OAE07 | Summary of All T-Cell Related Adverse Events by Maximum Grade | ICH E3 Use Combined PT list | SAC |
| 3.080 | mITT | OAE07 | Summary of All Lymphodepletion-Related Adverse Events by Maximum Grade | ICH E3 Use Combined PT list | SAC |
| 3.090 | ITT | AE15 | Summary of All Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) | FDAAA, EudraCT<br>Do not combine PT Terms | SAC |
| 3.100 | mITT | AE3 | Summary of All Non-Serious Study-Treatment Related AEs by Overall Frequency | Do not combine PT Terms | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events of Sp | ecial Interest | | | |
| 3.110 | mITT | ESI1 | Summary of Characteristics of Cytokine Release Syndrome-<br>First Infusion | Use Focused Scope List Report for all subjects and for all subjects with event Report characteristics, outcome, number of occurrences and max grade Do not create if 1 or less people have event, default to listing Footnote – "Preferred terms identified in the Focused list are summarized" Exclude AEs after second lymphodepletion | SAC |
| 3.140 | mITT | ESI1 | Summary of Characteristics of Haematopoietic Cytopenias (Comprehensive List)-First Infusion | Use Comprehensive Scope List Footnote – "Preferred terms identified in the Comprehensive list are summarized " See above | SAC |
| 3.180 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Cytokine Release Syndrome-First Infusion | Time to onset (days) (-81, 1-14, 15- 28, 29-56, >56) Remove subject at risk Duration (days) (1-28, 29-90, >90) Onset from first T-cell infusion Do not create if 1 or less people have event, default to listing Focused Scope reporting list Footnote – "Preferred terms identified in the Focused list are summarized | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.210 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Comprehensive List)-First Infusion | See note above- use comprehensive list Footnote – "Preferred terms identified in the Comprehensive list are summarized | SAC |
| 3.270 | mITT | ESI2a | Summary of Onset and Duration of the Last Occurrence of Haematopoietic Cytopenias (Comprehensive List)-First Infusion | See note above- use comprehensive list Footnote – "Preferred terms identified in the Comprehensive list are summarized | SAC |
| 3.290 | mITT | SAFE_T1 | Summary of Time to Resolution of Grade 3 and Above Cytokine Release Syndrome-First Infusion | Do not create if 1 or less people have event, default to listing Focused list | SAC |
| 3.320 | mITT | SAFE_T1 | Summary of Time to Resolution of Grade 3 and Above Haematopoietic Cytopenias (Comprehensive List)-First Infusion | Do not create if 1 or less people have event, default to listing | SAC |
| 3.360 | mITT | OAE01 | Summary of All Treatment Emergent Adverse Event of Special Interest by Maximum Grade (Focused List)-All Infusions | Replace SOC with AESI category Use Combined PT | SAC |
| 3.370 | mITT | OAE01 | Summary of All Treatment Emergent Adverse Event of Special Interest by Maximum Grade (Comprehensive List)-All Infusions | Replace SOC with AESI category Use preferred term, not combined PT | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 3.380 | ITT | AE16 | Summary of All Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT<br>Do not use Combined PT term | SAC |
| 3.390 | ITT | OAE07 | Summary of All Serious Adverse Events by Maximum Grade | Use Combined PT | SAC |
| 3.400 | mITT | OAE07 | Summary of All Treatment Emergent Serious Adverse Events by Maximum Grade | Use Combined PT | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.410 | mITT | OAE07 | Summary of All Study Treatment Related Serious Adverse Events by Maximum Grade | Use Combined PT Treatment related including all lymphodepletion regimens and T-cell Infusion | SAC |
| 3.420 | mITT | OAE07 | Summary of All T-cell Related Serious Adverse Events by Maximum Grade | Use Combined PT | SAC |
| 3.430 | mITT | OAE07 | Summary of All Lymphodepletion-Related Serious Adverse Events by Maximum Grade | Use Combined PT | SAC |
| 3.440 | ITT | AE3 | Summary of Fatal Adverse Events | Use Combined PT Don't produce if <5 subjects have fatal AE | SAC |
| 3.450 | mITT | AE3 | Summary of Study-Treatment Related Fatal Adverse Events | Don't produce if < 5 subjects have study treatment related fatal AE Use Combined PT | SAC |
| 3.460 | mITT | AE3 | Summary of All Serious Study-Treatment Related AEs by Overall Frequency | Don't use Combined PT | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Deaths | | | | | |
| 3.470 | mITT | DD1 | Summary of Deaths | IDSL Only report Alive at Last Contact, not follow up ended/ongoing Report as collected on the CRF -Disease Under study -Treatment related toxicity -Other Report time from T-cell infusion to death with median, min, max, 1st Q, 3rd Q in months, >30 days or <=30 days | SAC |
| Labora | tory: Chemistr | у | | | |
| 3.480 | mITT | LB1 | Summary of Chemistry Changes from Baseline (First Infusion) | ICH E3 | SAC |
| 3.490 | mITT | OBL9A | Summary of Worst Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline (First Infusion) | ICH E3 Do not report by visit For labs that are gradeable by CTCAEv4.03 | SAC |
| 3.500 | mITT | OLB11A | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline (First Infusion) | ICH E3 Do not report by visit For labs that are not gradeable by CTCAE | SAC |
| Labora | tory: Hematolo | уду | | | |
| 3.510 | mITT | LB1 | Summary of Hematology Changes from Baseline (First Infusion) | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.520 | mITT | OBL9A | Summary of Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline (First Infusion) | ICH E3 Do not report by visit For labs that are gradeable by CTCAEv4.03 | SAC |
| 3.530 | mITT | OLB11A | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline (First Infusion) | ICH E3 Do not report by visit For labs that are not gradeable by CTCAE | SAC |
| Labora | tory: Other Tes | sts | | | |
| 3.540 | mITT | LB1 | Summary of Urinalysis Laboratory Changes from Baseline (First Infusion) | ICH E3 | SAC |
| ECG | | | | | |
| 3.570 | mITT | EG1 | Summary of ECG Findings (First Infusion) | IDSL "Clinically significant change from baseline" in this standard shell is not collected in this study so cannot be reported: drop from display. | SAC |
| 3.580 | mITT | OECG1A | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (First Infusion) | IDSL Do not report by visit QTcF and QTcB reported in one table | SAC |
| 3.590 | mITT | EG2 | Summary of Change from Baseline in ECG Values by Visit (First Infusion) | IDSL<br>QTcF and QTcB reported separately | SAC |
| 3.600 | mITT | OECG2A | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category (First Infusion) | IDSL Do not report by visit QTcF and QTcB in one table | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 3.610 | mITT | VS1 | Summary of Change from Baseline in Vital Signs (First Infusion) | ICH E3 Include weight, bmi, temp, BP, pulse rate, respiratory rate, oxygen saturation | SAC |
| 3.620 | mITT | OVT1A | Summary of Worst Case change in Heart Rate Relative to Normal Range Post-Baseline Relative to Baseline (First Infusion) | IDSL Do not summarize by visit | SAC |
| 3.630 | mITT | OVT2A | Summary of Worst Case Increase in Blood Pressure by Maximum Grade Increase Post-Baseline Relative to Baseline (First Infusion) | IDSL Do not summarize by visit | SAC |
| Perforn | nance Status | | | | |
| 3.640 | mITT | PS1A | Summary of ECOG Performance Status (First Infusion) | ICH E3 Just summarize at baseline and last- assessment | SAC |
| 3.650 | mITT | PS3A | Summary of Change in ECOG Performance Status from Baseline (First Infusion) | ICH E3 Include best and worst case | SAC |
| Replica | tion Competer | nt Lentivirus Posi | tive (RCL) | | |
| 3.660 | mITT | SAFE_T3 | Summary of Replication Competent Lentivirus Positive | All infusions | SAC |
| 3.670 | mITT | SAFE_T3 | Summary of Subjects Showing >1% Gene Marked PBMCs 1<br>Year Post-treatment | Label- >1% Gene Marked PBMCs 1<br>Year Post-treatment<br>All infusions | SAC |

208749

## 14.10.8. Safety Figures

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Duratio | n Plots | | | | |
| 3.010. | mITT | SAFE_F1 | Plot of Prior Therapy Information | | SAC |
| 3.020. | mITT | SAFE_F2 | Plot of Duration on Interventional Phase 1 | | SAC |
| Laborat | tory | | | | |
| 3.030. | mITT | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT (First Infusion) | IDSL | SAC |
| 3.040. | mITT | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – eDISH (First Infusion) | IDSL | SAC |

## 14.10.9. Biomarker Tables

| Biomar | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Persist | ence of NY-ES | O-1 <sup>c259</sup> T | | | |
| 6.040 | mITT | | | Only report maximum persistence (i.e. not by scheduled visits). | 040 |
| 6.010. | | Report over | Report overall cohort and by responders vs. non-responders | SAC | |
| 6.020. | mITT | BIO_T2 | Summary of Time to Peak Persistence (First Infusion) | Report overall cohort and by responders vs. non-responders | SAC |

208749

## 14.10.10. Biomarker Figures

| Biomar | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Cytokir | nes | | | | |
| 6.010. | mITT | BIO_F4 | Profile of IL-6 by CRS Status and Subject (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Make CRS start red triangle, make CRS stop red square. Add legend labels for start and stop of CRS event. Add label of CRS start and stop date Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.020. | mITT | BIO_F4 | Profile of IL-6 by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.030. | mITT2 | BIO_F4 | Profile of IL-6 by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use Log10 for y axis and same x axis length as first infusion display | SAC |

| Biomar | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.040. | mITT | BIO_F4 | Profile of IL-10 by CRS Status and Subject (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Make CRS start red triangle, make CRS stop red square. Add legend labels for start and stop of CRS event. Add label of CRS start and stop date Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.050. | mITT | BIO_F4 | Profile of IL-10 by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.060. | mITT2 | BIO_F4 | Profile of IL-10 by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use Log10 for y axis and same x axis length as first infusion display | SAC |
| 6.070. | mITT | BIO_F4 | Profile of TNF-alpha by CRS Status and Subject (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Make CRS start red triangle, make CRS stop red square. Add legend labels for start and stop of CRS event. Add label of CRS start and stop date Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |

| Biomar | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.080. | mITT | BIO_F4 | Profile of TNF-alpha by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.090. | mITT2 | BIO_F4 | Profile of TNF-alpha by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use Log10 for y axis and same x axis length as first infusion display | SAC |
| 6.100. | mITT | BIO_F4 | Profile of IFN-gamma by CRS Status and Subject (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Make CRS start red triangle, make CRS stop red square. Add legend labels for start and stop of CRS event. Add label of CRS start and stop date Add dot at each cytokine measurement One color per subject Use Log10 for y axis | SAC |
| 6.110. | mlTT | BIO_F4 | Profile of IFN-gamma by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject Use Log10 for y axis. | SAC |

| Biomar | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.120. | mITT2 | BIO_F4 | Profile of IFN-gamma by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use Log10 for y axis and same x axis length as first infusion display | SAC |
| 6.130. | mITT | BIO_F4 | Profile of IL-1beta by CRS Status and Subject (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Make CRS start red triangle, make CRS stop red square. Add legend labels for start and stop of CRS event. Add label of CRS start and stop date Add dot at each cytokine measurement One color per subject | SAC |
| 6.140. | mlTT | BIO_F4 | Profile of IL-1beta by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject | SAC |
| 6.150. | mITT2 | BIO_F4 | Profile of IL-1beta by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use same x axis length as first infusion display | SAC |
| 6.151 | mITT | BIO_F4 | Profile of IL-7 by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject | SAC |

| Biomar | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.152 | mITT2 | BIO_F4 | Profile of IL-7 by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use same x axis length as first infusion display | SAC |
| 6.153 | mITT | BIO_F4 | Profile of IL-15 by Response and Subject (First Infusion) | By responder and non-responder per investigator-assessed best response with confirmation. Include footnote per mock programming note. Add dot at each cytokine measurement One color per subject | SAC |
| 6.154 | mITT2 | BIO_F4 | Profile of IL-15 by Subject (Second Infusion) | Do not separate by responder status Add dot at each cytokine measurement Use same x axis length as first infusion display | SAC |
| 6.160. | mITT | BIO_F5 | Peak Cytokine Expression of IL-6 by CRS Status (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Add mean in legend | SAC |
| 6.170. | mITT | BIO_F5 | Peak Cytokine Expression of IL-6 by Response (First Infusion) | By responder and non-responder Add mean in legend | SAC |
| 6.180. | mITT | BIO_F5 | Peak Cytokine Expression of IL-10 by CRS Status (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Add mean in legend | SAC |
| 6.190. | mITT | BIO_F5 | Peak Cytokine Expression of IL-10 by Response (First Infusion) | By responder and non-responder<br>Add mean in legend | SAC |
| 6.200. | mITT | BIO_F5 | Peak Cytokine Expression of TNF-alpha by CRS Status (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Add mean in legend | SAC |

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.210. | mITT | BIO_F5 | Peak Cytokine Expression of TNF-alpha by Response (First Infusion) | By responder and non-responder Add mean in legend | SAC |
| 6.220. | mITT | BIO_F5 | Peak Cytokine Expression of IFN-gamma by CRS Status (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Add mean in legend | SAC |
| 6.230. | mITT | BIO_F5 | Peak Cytokine Expression of IFN-gamma by Response (First Infusion) | By responder and non-responder<br>Add mean in legend | SAC |
| 6.240. | mITT | BIO_F5 | Peak Cytokine Expression of IL-1beta by CRS Status (First Infusion) | By CRS (None or Non-Serious CRS vs. Serious CRS) Add mean in legend | SAC |
| 6.250. | mITT | BIO_F5 | Peak Cytokine Expression of IL-1beta by Response (First Infusion) | By responder and non-responder Add mean in legend | SAC |
| 6.251 | mITT | BIO_F5 | Peak Cytokine Expression of IL-7 by Response (First Infusion) | By responder and non-responder Add mean in legend | SAC |
| 6.252 | mITT | BIO_F5 | Peak Cytokine Expression of IL-15 by Response (First Infusion) | By responder and non-responder<br>Add mean in legend | SAC |
| Persist | ence of NY-ES | O-1 <sup>c259</sup> T | | | |
| 6.260. | mITT | BIO_F3 | Persistence Profile by Subject (First Infusion) | Do not separate responder and non-<br>responder Create a new display for each subject All subjects should not be on the same<br>plot. Use same x and y axis for all plots | SAC |
| 6.270. | mITT | BIO_F3 | Persistence Profile by Subject and Responder Status (First Infusion) | Separate by responder and non-<br>responder All subjects in the same display | SAC |

| Biomarker: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.271 | mITT | BIO_F3 | Persistence Profile by Subject and Responder Status<br>Truncated at 6 Months (First Infusion) | Separate by responder and non-<br>responder All subjects in the same display Truncate at day 180 and show tick mark every 30 days | SAC |
| 6.280. | mITT2 | BIO_F3 | Persistence Profile by Subject (Second Infusion) | Do not separate by responder-non-responder Use x axis length in display 6.260 | SAC |
| 6.290. | mITT | BIO_F5 | Distribution of Peak Persistence (First Infusion) | By responder and non-responder<br>Add mean in legend | SAC |

208749

## 14.10.11. ICH Listings

Add mITT and mITT2 flags to all ITT listings and mITT2 flags to all mITT listings. Replace Study Day in all listings to Time from 1st Infusion/ Time from 2nd Infusion

| ICH: Listin | gs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Subject Di | sposition | | | | |
| 10. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines Only include subjects that were screen failures Do not include "Type of Failure" | SAC |
| 20. | ITT | ES2 | Listing of Reasons for Study Withdrawal (Interventional Phase 1) | ICH E3 Do not include columns "Reason Term(s)", "Was a follow-up phone contact attempted 3 times?" & "Was a follow-up certified letter mailed?" from GSK standard mock as not collected in this study. | SAC |
| 30. | Second T-<br>cell<br>Infusion | ES2 | Listing of Reasons for Study Withdrawal (Interventional Phase 2) | ICH E3Do not include columns "Reason Term(s)", "Was a follow-up phone contact attempted 3 times?" & " Was a follow-up certified letter mailed?" from GSK standard mock as not collected in this study. | SAC |
| 40. | mITT | POP_L5 | Listing of Subject Status | | SAC |
| Protocol D | eviations | | | | |
| 50. | ITT | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 60. | ITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |

| ICH: Listing | gs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Population | s Analysed | | | | • |
| 70. | Screened | SP3 | Listing of Subjects Excluded from Any Population | ICH E3<br>ITT, mITT, mITT2 | SAC |
| Demograpl | hic and Baselii | ne Characteristics | | | |
| 80. | ITT | DM2 | Listing of Demographic Characteristics | ICH E3<br>Add BMI and Race | SAC |
| Prior and C | Concomitant M | edications | | | |
| 90. | ITT | BP4 | Listing of Blood Products | IDSL Include flag for blood product occurring on or after second lymphodepletion | SAC |
| 100. | ITT | CM3 | Listing of Medications | IDSL Include all collected medications, do not subset on concomitant medications study phase Replace "Started Pre-Trial" column with "Prior / Concomitant" Include flag for conmed occurring on or after second lymphodepletion | SAC |
| Exposure a | and Treatment | Compliance | | | • |
| 110. | ITT | Non-standard/POP_L3 | Listing of Leukapheresis, Lymphodepletion, and T-cell Infusion Dates | ICH E3 Include both first and second infusion exposures | SAC |

| ICH: Listing | js | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 120. | ITT | POP_L1 | Listing of Exposure to T-cell Infusion | ICH E3 Start date, study day, start time, end time, total cell dose, total number of transduced cells, percentage of cells transduced, lot number. Report cell dose as 10^9 Include both first and second infusion exposures | SAC |
| 130. | ITT | POP_L2 | Listing of Exposure to Lymphodepletion Chemotherapy | ICH E3 Include both first and second infusion exposures | SAC |
| Response | | | | | |
| 140. | ITT | RE5 | Listing of Investigator-Assessed Responses at Each Visit with Confirmation (RECIST 1.1 Criteria)- First Infusion | Include Target and Non-Target Lesion column Do not keep measureable disease at baseline ,CA, or organs of PD columns Include footnote identify subject that does not have target lesion at baseline | SAC |
| 150. | mITT2 | RE5 | Listing of Investigator-Assessed Responses at Each Visit with Confirmation (RECIST 1.1 Criteria)- Second Infusion | Include Target and Non-Target Lesion column Do not keep measureable disease at baseline ,CA, or organs of PD columns | SAC |
| 160. | mITT | TTE9 | Listing of Time To Response -First Infusion | Change randomization date to T-cell Infusion Date, | SAC |

| ICH: Listing | gs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 170. | mITT | TTE9 | Listing of Time To Response -Second Infusion | Change randomization date to 2nd T-cell Infusion Date, | SAC |
| 180. | mITT | TTE9 | Listing of Progression-Free Survival-First Infusion | Use T-cell infusion date Include footnote identify subject that does not have target lesion at baseline | SAC |
| 190. | mITT | TTE9 | Listing of Progression-Free Survival-Second Infusion | Use T-cell infusion date | SAC |
| 200. | mITT | TTE9 | Listing of Duration of Response-First Infusion | Change randomization date to T-<br>cell Infusion Date. Add date of<br>confirmed response | SAC |
| 210. | mITT | TTE9 | Listing of Duration of Response-Second Infusion | Change randomization date to 2nd T-cell Infusion Date. Add date of confirmed response | SAC |
| 220. | mITT | TTE9 | Listing of Overall Survival | Change randomization date to T-cell Infusion Date. | SAC |
| Adverse Ev | vents | | | | |
| 230. | ITT | AE8 | Listing of Adverse Events | ICH E3 Use "Time Since 1st T-Cell Infusion/Time Since 2nd T-cell Infusion" MITT flag Include all AEs on study and display flag for second infusion treatment emergent AE (Y/N) | SAC |

| ICH: Listing | js | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 240. | mITT | SAFE_L1 | Listing of Delayed Adverse Events | ICH E3 Use "Time Since 1st T-Cell Infusion/Time Since 2nd T-cell Infusion" Display second infusion treatment emergent AE flag | SAC |
| 250. | ITT | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3<br>All AEs | SAC |
| 260. | ITT | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Adverse Ev | ents of Specia | al Interest | | | |
| 270. | mITT | SAFE_L1 | Listing of Cytokine Release Syndrome Adverse Events | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 Add column Medications/Procedures | SAC |
| 280. | mITT | SAFE_L2 | Listing of Symptoms, Concomitant Medications, and Procedures Related to Cytokine Release Syndrome | | SAC |
| 290. | mITT | SAFE_L1 | Listing of Graft versus Host Disease Adverse Events | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |

| ICH: Listing | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 300. | mITT | SAFE_L1 | Listing of Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS)- Adverse Events | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |
| 310. | mITT | SAFE_L1 | Listing of Haematopoietic Cytopenias Adverse Events (Focused List) | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |
| 320. | mITT | SAFE_L1 | Listing of Haematopoietic Cytopenias Adverse Events (Comprehensive List) | Comprehensive scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |
| 330. | mITT | SAFE_L1 | Listing of Guillain-Barre Syndrome Adverse Events | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |
| 340. | mITT | SAFE_L1 | Listing of Pneumonitis Adverse Events | Focused scope Sort by USUBJID, AEDECOD, ASTDT, AENDT Display all AESIs, 1st and 2nd inf. Display start and end study day 2 | SAC |

| ICH: Listing | gs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious and | d Other Signif | icant Adverse Events | | | |
| 350. | ITT | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 Use "Time Since 1st T-Cell Infusion/Time Since 2nd T-cell Infusion" Display all AEs MITT Flag Display second infusion treatment emergent AE flag | SAC |
| 360. | ITT | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 Use "Time Since 1st T-Cell Infusion/Time Since 2nd T-cell Infusion" MITT Flag Display all AEs Display second infusion treatment emergent AE flag | SAC |
| 370. | ITT | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 Display second infusion treatment emergent AE flag | SAC |
| 371. | ITT | PAN12 | Listing of Covid-19 Assessments and Symptoms Assessments | If data exists | SAC |

| ICH: Listing | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Deaths | | | | · | |
| 380. | ITT | DTH3 | Listing of Deaths | ICH E3 Include "Time from 1st T-cell infusion/ Time from 2nd T-cell infusion" MITT Flag Exclude "No. of Cycles/ Last Dose (unit)". | SAC |
| 381 | ITT | DD3 | Death Profile | ICH E3 MITT Flag If data warrant | SAC |
| Hepatobilia | ry (Liver) | | | · | |
| 390. | ITT | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL Update columns "Time Since First Dose", "Time Since Last Dose (days)" of LIVER5 mock with "Time Since First T-Cell Infusion" & "Time Since Second T-Cell Infusion". | SAC |
| 400. | mITT | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory Criteria Post-Baseline | IDSL | SAC |
| 410. | ITT | LIVER15 | Liver Stopping Event Profile | IDSL Date of Start of Treatment and Date of End of Treatment change to Date of First T-cell Infusion, Date of Second T-cell Infusion | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Laborat | tory | | | | 1 |
| 420. | ITT | LB5A | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC |
| 430. | ITT | LB5A | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC |
| 440. | ITT | LB5A | Listing of All Other Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC |
| 450. | ITT | LB5A | Listing of Chemistry Values of Potential Clinical Importance | | SAC |
| 460. | ITT | LB5A | Listing of Hematology Values of Potential Clinical Importance | | SAC |
| 470. | ITT | LB5A | Listing of Other Laboratory Values of Potential Clinical Importance | | SAC |
| 480. | ITT | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 490. | ITT | UR2A | Listing of Urinalysis Data | ICH E3 | SAC |
| 500. | mITT | LB5 | Listing of Cytokine Data | Include flag for subjects with serious CRS event Include all infusions | SAC |
| 510. | mITT | BIO_L1 | Listing of Persistence Data | Raw and Derived All infusions included with second infusion info derived separately | SAC |
| 520. | mITT | LB5 | Listing of VSV-G DNA (RCL) Data | | SAC |
| 531. | mITT | LB5 | Listing of ICE Score | Date, Time, ICE Points | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 532. | ITT | BIO_L2 | Listing of Immunohistochemistry Data | | SAC |
| ECG | | | | | |
| 540. | ITT | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 550. | ITT | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL Remove clinically significant change from baseline and clinically significant abnormality | SAC |
| 560. | ITT | OECG5A | Listing of QTc Values of Potential Clinical Importance | Specify if Bazett's or Fridericia | SAC |
| Vital Signs | | | | | |
| 570. | ITT | OVT7A | Listing of Vital Signs with any Value of Potential Clinical Importance | Add oxygen saturation column with category defined in PCI section | SAC |
| Performance Status | | | | | |
| 580. | ITT | PS5A | Listing of ECOG Performance Status | | SAC |
208749

# 14.10.12. Non-ICH Listings

Add mITT and mITT2 flags to all ITT listings and mITT2 flags to all mITT listings

| Non-ICH: Lis | Sungs | IDSL / | | | |
|---|---|---|---|---|---|
| No. | Population | Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Disease Cha | racteristics | | | | |
| 590. | ITT | DC3 | Listing of Disease Characteristics at Initial Diagnosis | Date of diagnosis/ time from diagnosis to screening (months), stage of lung cancer at initial diagnosis, type of histology | SAC |
| 600. | ITT | POP_L4 | Listing of Disease Characteristics at Screening | Number of prior systemic therapy regimens before enrolment, number of radiotherapy therapy before enrolment,*, stage of lung cancer at time of enrolment, Tumor Type, Anatomical Location, HLA Allele 1 status, HLA Allele 2 status, NY-ESO-1 status | SAC |
| Anti-Cancer | Therapy | | | | |
| 610. | ITT | AC6 | Listing of Prior Anti-Cancer Therapy | Include amount/scheduled or cumulative dose, regimen number, and best response per mock Therapy before leukapheresis-see study phase | SAC |
| 611. | ITT | AC6 | Listing of Bridging Anti-Cancer Therapy | Include amount/scheduled or cumulative dose and regimen number, and best response per mock | SAC |

208749

| No. Population Example Shell | | Example | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | see study phase for definition of bridging therapy | |
| 620. | mITT | FAC3 | Listing of On-Study Anti-Cancer Therapy | Include flag for on-study anti-cancer therapy occurring on or after second lymphodepletion Include amount/scheduled or cumulative dose and regimen number per mock | SAC |
| 630. | ITT | AC7 | Listing of Prior and Bridging Anti-Cancer Radiotherapy | Include prior and bridging and flag bridging therapy | SAC |
| Medical Cor | nditions | | | | |
| 640. | ITT | MH2 | Listing of Medical Conditions | Remove Past/Current category and replace with "Ongoing?" flag | SAC |
| Surgical Pro | ocedures | | | | |
| 650. | ITT | OSP3 | Listing of Prior and Bridging Cancer-Related Surgical Procedures | List Surgery Intent and Site and Date of Surgery Include prior and bridging and flag bridging therapy | SAC |
| 660. | mITT | OSP3 | Listing of On-Study Cancer-Related Surgical Procedures | List Surgery Intent and Site and Date of Surgery Include flag for on-study surgery occurring on or after second lymphodepletion | SAC |
| 661. | ITT | OSP3 | Listing of Tumor Biopsies | Use listing 650 as mock and remove timepoint, classification, and bridging therapy column. Rename "Surgery Intent"="Type of Sample Obtained", "Site of Surgery" | SAC |

208749

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | = "Anatomical Location" | |
| Substance Us | Substance Use | | | | |
| 670. | ITT | SU2 | Listing of Substance Use | List cigarette use, years smoked, packs per day | SAC |
| Responses | Responses | | | | |
| 680. | mITT | LA5 | Listing of Investigator-Assessed Lesion Assessments (RECIST 1.1 Criteria) | Include second infusion lesion assessments | SAC |

208749

#### 14.11. **Appendix 11: Example Mock Shells for Data Displays**

# 14.11.1. POP\_T1 Exposure Mock-Up Summary

Example POP T1

Protocol: 208479  Population: Intent-To-Treat

(Data as of: 24APR2018)

GSK794

Table X.X Summary of Exposure

| | (N=15) |
|----------------------------------|----------|
| Apheresis Performed | 13 (87%) |
| Received Lymphodepleting Therapy | 12 (80%) |
| Received T-cell Infusion | 10 (67%) |
| Received Second T-cell Infusion | 2 (13%) |

#### Note:

<sup>1:</sup> ITT population comprises of all subjects who enrolled in the trial and met all eligibility criteria.. PPD

208749

# 14.11.2. EFF\_F1 Spider Plot Mock-Up Figure

Example EFF\_F1

Protocol: 208479 
Population: Modified Intent-to-Treat (Data as of: 24APR2018)

Figure X
Spider Plot of Percent Change from Baseline in Target Lesion Diameter



#### Note:

1: mITT population includes all ITT subjects who received T cell infusion.

# 14.11.3. SAFE\_F1 Prior Therapy Mock-Up Figure

Figure 1.15
Plot of Prior Therapy Information



# 14.11.4. SAFE\_F2 Study Duration Mock Up Figure



208749

208749

#### 14.11.5. **BIO\_F3 Persistence Profile Mock-Up Figure**

Example BIO F3

Protocol: 208479  (Data as of: 24APR2018)

Population: Modified Intent-to-Treat

Figure X





Note 1: mITT (modified Intent to Treat) is defined as all eligible subjects who received T-Cell therapy Note 2: Y axis is Log Transformed. Values that are <xx are set to 1.

Source: P:\Biometrics\05Sep2017Datacutoff\04511\Programs\perplt\_coh1.sas Run Date\Time: 10/18/2017 16:03

#### Note:

1: mITT population includes all ITT subjects who received T cell infusion.

208749

# 14.11.6. BIO\_F4 Cytokine Spider Plot Mock-Up Figure

Example BIO\_F4
Protocol: 208479

Population: Modified Intent-to-Treat

 (Data as of: 24APR2018)

Figure X IL-6 Profile by Subject



#### Note:

1: mITT population includes all ITT subjects who received T cell infusion
Where plotting split by responder and non-responder include footnote "Note: Responders are subjects with investigator-assessed best response with confirmation (per RECIST 1.1 criteria) of Partial Response or Complete Response."

208749

# 14.11.7. BIO\_F5 Cytokine Box Plot Figure

Example BIO\_F5
Protocol: 208479

Population: Modified Intent-to-Treat

 (Data as of: 24APR2018)





#### Note:

1: mITT population includes all ITT subjects who received T cell infusion

208749

# 14.11.8. SAFE\_L1 CRS Mock-Up Listing

Example SAFE\_L1
Protocol: GSK208479

Protocol: GSK208479

Population: Intent-to-Treat

Page 1 of n

(Data as of: 24APR2018)

Listing XX

Listing of Adverse Events of Special Interest

Treatment: GSK794

Infusion: First Infusion

| Site Id./<br>Unique<br>Subject Id. | Date of Apheresis/ Date of Lymphodepletio n/ Date of T-cell Infusion | Preferre<br>d Term | Event | AE Start Date/Star t Study Day/ AE End Date/End Study Day/ Event Duration (Days) | SAE Code | Grad<br>e | Relationshi<br>p to Study<br>Treatment | Outcome of Event |
|---|---|---|---|---|---|---|---|---|
| PPD /<br>PPD | PPD / | Cytokine<br>release<br>syndrome | 9 | PPD<br>/ 3<br>PPD<br>/ 10/<br>8 | Not applicab | le Grad<br>e 2 | Yes: T-<br>Cell | Recovered/resolv ed |
| | | | | PPD / 5 PPD / 11 7 | Not applicab | le Grad<br>e 3 | Yes: T-<br>Cell | Recovered/resolv ed |

208749



#### Note:

- 1: ITT population comprises of all subjects who enrolled in the trial and met all eligibility criteria.
- 2: The second infusion section of the listing includes all AE starting after second lymphodepletion. In the section, the study day is in reference to second T-cell infusion, and the apheresis, lymphodepletion, and T-cell dates are for second infusion.

USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.9. BIO\_T1 Summary of Peak Persistence

Example BIO T1

Protocol: 208749  (Data as of: 24APR2018)

Population: Modified Intent-to-Treat

Table X Summary of Peak Persistence

| Test (units) | Group | N | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| Peak Persistence<br>(Cell number/ µL) | Overall | 202 | 180 | 74.3 | 9.82 | 74 | 51 | 96 |
| | Non-<br>Responders | 100 | 90 | 70.4 | 8.51 | 62 | 51 | 80.4 |
| | Responders | 102 | 90 | 80.4 | 6.41 | 92 | 30 | 96 |

#### Note:

<sup>1:</sup> mITT population comprises of all subjects in the ITT population that received T-cell infusion PPD

208749

# 14.11.10. BIO\_T2 Summary of Time to Peak Persistence

Example: BIO\_T2

Protocol: 208749 
Population: Modified Intent-to-Treat (Data as of: 24APR2018)

Time (Days) to Peak Persistence (Cell number/  $\mu L$ ) Group Ν SD Median Min. Max. n Mean 99 25.0 4.52 25.0 20 34 Overall 100 3.25 22.0 Non-Responders 20 28 21.0 50 49 Responders 50 50 30.0 3.51 29.5 36 34

#### Note:

1: mITT population comprises of all subjects in the ITT population that received T-cell infusion PPD

208749

# 14.11.11. SAFE\_T3 Summary of Replication Competent Lentivirus Positive

Example: BIO\_T3

Protocol: 208749 
Population: Modified Intent-to-Treat (Data as of: 24APR2018)

| | GSK794<br>(N=40) |
|-------------------------------------------|------------------|
| Replication Competent Lentivirus Positive | |
| n | 4 |
| Count | 2 (50%) |

#### Note:

1: mITT population comprises of all subjects in the ITT population that received T-cell infusion PPD

208749

# 14.11.12. BIO\_L1 Listing of Persistence

Example: BIO\_L1

Listing of Persistence Results

Treatment=Treatment A

| Site<br>ID/Subject ID | Age<br>(YEARS<br>)/<br>Sex/<br>Race | Planne<br>d<br>Time | Date/Stu<br>dy Day | / Number | Copie<br>s per<br>Cell/<br>Perce<br>nt<br>gene<br>marke<br>d<br>PBMCs<br>(%) | Copes<br>per<br>ug<br>DNA | Interpreti<br>ve<br>Result | Peak Persistenc e/ Time to Peak Persistenc e (days) | Time to 25% Loss of Peak Persistence (days)/50%/7 5%/ Duration of Detectable Persistence |
|---|---|---|---|---|---|---|---|---|---|
| PPD /<br>PPD | 65/<br>F/<br>MULTIP<br>LE | Baseli<br>ne | PPD -11 | N/A/<br>1 | <.000<br>3/<br>0% | <50.0 | NEGATIVE | 67852.7/<br>2 | 3/<br>14/<br>14/<br>28+ |
| | | Day 1 | PPD / 1 | N/A/<br>1 | <.001<br>6 | <250.<br>0 | NEGATIVE | | |
| | | Day 2 | PPD<br>PPD/ 2 | .2/ | .4275<br>/<br>42.75<br>% | 67852 | POSITIVE | | |

| Day 4 | PPD<br>PP / 4 | .1/ | .2544<br>/<br>25.44<br>% | 40383 | POSITIVE |
|---|---|---|---|---|---|
| Day 8 | PPD PP / 8 | .2/ | .4226<br>/<br>42.26<br>% | 67080<br>.7 | POSITIVE |
| Week 2 | PPD PP / 14 | .3/ | .0173<br>/<br>1.73% | 2742.<br>5 | POSITIVE |
| Week 4 | PPD | .2/<br>28 | .0041<br>/<br>.41% | 644.2 | POSITIVE |

208749

# 14.11.13. POP\_L1 Listing of Exposure to T-cell Infusion

Example: POP\_L1 Protocol: 208749

Protocol: 208749 
Population: Intent-to-Treat (Data as of: 24APR2018)

Listing X
Listing of Exposure to T-cell Infusion

Treatment: GSK794

| Centre Id./ Subject | Start<br>Date/Start<br>Time/<br>Study Day | Stop<br>Date/Stop<br>Time/<br>Study Day | Total Number of Transduced Cells (10^9 cells) | Percentage of Cells Transduced (%) |
|---|---|---|---|---|
| PPD / | PPD /<br>14:30/<br>1 | PPD /<br>15:30/<br>1 | 1.21 | 35.4 |
| PPD / | PPD / 10:30/ | PPD / | 2.52 | 28.3 |

#### Note:

1: ITT population comprises of all subjects who enrolled in the trial and met all eligibility criteria. USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.14. POP\_L2 Listing of Exposure to Cyclophosphamide/Mesna

Example: POP\_L2

Protocol: 208749 
Population: Intent-to-Treat (Data as of: 24APR2018)

Listing X

Listing of Exposure to Lymphodepletion Chemotherapy Medicine

Treatment: LOW LYMPHO DOSE + GSK794

| Centre A<br>Id./Uniq | Age Visit | Cyclophosphamide<br>Administration | e<br>Fludarabine Administration |
|---|---|---|---|
| ue<br>Subject | | Infusion Dose/Unit<br>Date/Study<br>Day | Infusion Dose/Unit Date/Study Day |
| PPD /<br>PPD | | <b>PPD</b> / -7 | <u>*</u> |

<sup>1:</sup> ITT population comprises of all participants who enrolled in the trial and met all eligibility criteria. USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.15. POP\_L3 Listing of Leukapheresis, Lymphodepletion, and T-cell Infusion Dates

Example: POP\_L3
Protocol: 208749

Population: Intent-to-Treat
(Data as of: 24APR2018)

Listing X

Listing of Leukapheresis, Lymphodepletion, and T-cell Infusion Dates

Treatment: GSK794

| Centre Id./<br>Subject | Visit | Treatment | Date /<br>Study Day |
|------------------------|-----------|------------------|---------------------|
| PPD /<br>PPD | Screening | APHERESIS | <b>PPD</b> / -60 |
| | | FLUDARABINE | <b>PPD</b> / -8 |
| | | FLUDARABINE | <b>PPD</b> / -7 |
| | | CYCLOPHOSPHAMIDE | PPD / -7 |
| | | MESNA | PPD / -7 |
| | | FLUDARABINE | <b>PPD</b> / -6 |

208749

| CYCLOPHOSPHAMIDE | <b>PPD</b> / -6 |
|------------------|-----------------|
| MESNA | <b>PPD</b> / -6 |
| FLUDARABINE | <b>PPD</b> / -5 |
| CYCLOPHOSPHAMIDE | <b>PPD</b> / -5 |
| MESNA | <b>PPD</b> / -5 |
| T-CELL | PPD / 1 |

#### Note:

1: ITT population comprises of all subjects who enrolled in the trial and met all eligibility criteria. USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.16. POP\_L4 Listing of Disease Characteristics at Screening

Example: POP\_L4
Protocol: 208749

Protocol: 208749 
Population: Intent-to-Treat (Data as of: 24APR2018)

Listing X

Listing of Disease Characteristics at Screening

Treatment: GSK794

| Centre<br>Id./<br>Subject | Number of<br>Prior Anti-<br>Cancer<br>Therapy<br>Regimens[1] | Cancer at<br>Time of | Tumor Type | Anatomical<br>Location | Date of<br>Blood<br>Collection<br>for HLA<br>Testing | HLA Allele | HLA Allele 2 | Date of<br>Biopsy<br>for<br>Antigen<br>Testing | NY-ESO-1<br>Status |
|---|---|---|---|---|---|---|---|---|---|
| PPD / | 2 | STAGE IIIB | METASTATIC | LUNG | PPD | HLA-<br>A*02:01 | OTHER, NOT<br>HLA-A*02 | PPD | POSITIVE |
| PPD / | 3 | STAGE 4 | PRIMARY | LUNG | PPD | HLA-<br>A*02:01 | HLA-A*02:01 | PPD | NEGATIVE |

#### Note:

1: Number of regimens includes all regimens before start of lymphodepleting chemotherapy USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.17. POP\_L5 Subject Status Mock-Up Listing

Example POP\_L5

Protocol: GSK208749 Page 1 of n

Population: Intent-to-Treat

Listing XX Listing of Subject Status

| Site Id./<br>Unique Subject<br>Id. | Lymphodepletion (Y/N) | 1st T Cell Infusion Date/Time between Leukapheresi s and 1st T- cell Infusion/ 2nd T Cell Infusion Date | 1st Transduce d Dose (10^9 cells)/ 2nd Transduce d Dose (10^9 cells) | Completed Interventiona l Phase 1/ 2 (Y/N) | Date of Discontinuatio n or Completion of Interventional Phase 1/ 2 | n or<br>Completion of | End of<br>Study<br>Reason |
|---|---|---|---|---|---|---|---|
| PPD /<br>PPD | Y | PPD / | 4.52/<br>3.24 | Y/<br>N | PPD / | Progressive<br>disease/<br>Death | Death |
| PPD /<br>PPD | Y | PPD | 6.24 | N | PPD | Withdrew<br>consent | Withdre<br>w<br>consent |

#### Note:

<sup>1:</sup> ITT population comprises of all subjects who enrolled in the trial and met all eligibility criteria..

208749

# 14.11.18. EFF\_T1 Summary of Time to Response by Investigator (RECIST 1.1 Criteria)

Example EFF\_T1

Protocol: 208749


Population: eq. Intent to Treat/Safety/Other Study Specific

Population: eg, Intent to Treat/Safety/Other Study Specific Table  ${\tt X}$ 

Summary of Time to Response by Investigator (RECIST 1.1 Criteria)

| | GSK749<br>(N=100) |
|---|---|
| Number of Subjects with Confirmed Response | 50/100 (50%) |
| Time to Response (months) Min 1st Quartile Median 3rd Quartile | 3<br>4.3<br>5.4<br>10.8 |
| Max. | 12 |

#### Note:

1: mITT population comprises of all subjects in the ITT population that received T-cell infusion PPD

208749

# 14.11.19. SAFE\_T1 Summary of Time to Resolution

SAFE T1

Table 3.5610

Summary of Time to Resolution of Grade 3 and Above Adverse Event of Special Interest - Haematopoietic Cytopenias (Comprehensive List - First Infusion)

| | | GSK749<br>(N=5) |
|---|---|---|
| Initial Occurence <= Study Day 28 | n | 4 |
| | <= Study Day 28<br>Study Day 29 - 90<br>Study Day >90<br>Unresolved | 4 (100%)<br>0<br>0 |
| Recurrence > Study Day 28 | n | 0 |
| | <= 28 Days<br>29 - 90 Days<br>>90 Days<br>Unresolved | 0<br>0<br>0 |

Segment 1: Any subject with events starting on or before Day 28 are considered for the first segment. Time to resolution in relation to T-cell infusion is being summarized

Ex: Subject with one AE starting on Study Day 27 that resolved on Study Day 29 will be summarized in the "Study Day 29-90" row.

Segment 2: Recurrent events starting after Day 28 for those subset of subjects in segment 1 Time to resolution in relation to overall duration of the event is summarized

If a subject has multiple events that fall within the time of interest, the worst case is summarized. Unresolved is worst case.

Modified Intent-to-Treat population includes all subjects who received T-cell infusion.

208749

# 14.11.20. POP\_T2 Summary of Subject Status

Example POP\_T2
Protocol: 208749

Protocol:  $2\overline{0}8749$  

Population: Intent-to-Treat (Data as of: 24APR2018)

# Table X.X Summary of Subject Status

| | GSK794 | (N=300) |
|------------------------------------------------|--------|----------|
| INTERVENTIONAL PHASE 1 STATUS | | |
| COMPLETED | XX (X | X%) |
| NOT PROGRESSED AT 2 YEARS POST T-CELL INFUSION | XX (X | · |
| PROGRESSIVE DISEASE | XX (X | ,<br>Х%) |
| DIED | XX (X | X%) |
| ONGOING | XX (X | X용) |
| DID NOT COMPLETE | XX (X | X%) |
| WITHDREW CONSENT | XX (X | X%) |
| FAILED TO MEET ELIGIBILITY PRIOR TO | XX (X | X%) |
| CYTOREDUCTIVE CHEMOTHERAPY | | |
| FAILED TO MEET ELIGIBILITY PRIOR TO | XX (X | X%) |
| LEUKAPHERESIS | | |
| LOST TO FOLLOW-UP | XX (X | X%) |
| INVESTIGATOR DISCRETINOY | XX (X | X%) |
| STUDY TERMINATED BY SPONSOR | XX (X | X%) |
| DID NOT RECEIVE T-CELL INFUSION | XX (X | X%) |
| DEATH (PRIOR TO T-CELL INFUSION) | XX (X | X%) |
| OTHER | XX (X | X%) |

208749

# 14.11.21. POP\_T3 Summary of Subject Status- End of Study

Example POP\_T2

Protocol: 208749 

Population: Intent-to-Treat (Data as of: 24APR2018)

Table X.X
Summary of Subject Status

DEATH XX (XX%)
WITHDREW CONSENT XX (XX%)
MOVED TO LTFU STUDY XX (XX%)
LOST TO FOLLOW-UP XX (XX%)
OTHER XX (XX%)

208749

# 14.11.22. SAFE\_L2 Listing of Symptoms, Concomitant Medications, and Procedures Related to Cytokine Release Syndrome

Example SAFE L2

Protocol: GSK208749 Page 1 of n
Population: Modified Intent-to-Treat (Data as of: 24APR2018)

Listing XX

Listing of Concomitant Medications and Procedures Related to Cytokine Release Syndrome

| Site Id./<br>Unique<br>Subject<br>Id. | Apheresis/<br>Date of<br>Lymphodepleti<br>on/ | Infusion/ Time from $2^{nd}$ T-cell | Symptoms | Medications | Procedures |
|---|---|---|---|---|---|
| PPD /<br>PPD | PPD / | <b>PPD</b> / 3/ | HYPOXIA, OTHER: ventricular tachycardia | IV FLUIDS,<br>OTHER:ACETAMINOPHEN | VENTILATION ASSISTANCE |
| PPD /<br>PPD | PPD / | <b>PPD</b> / 5/ | | CORTICOSTEROIDS, TOCILIZUMAB, OTHER: ACETAMINOPHEN | |
| PPD /<br>PPD | PPD | PPD / 5/ | | , POTASSIUM<br>CHLORIDE | OXYGEN |

 $\hbox{Note: Modified Intent-to-Treat (mITT) population includes all enrolled subjects who were dosed}\\$ 

Note: Medications and procedures as recorded on "CYTOKINE RELEASE SYNDROME" form.

USER ID:directory/program.sas 01JAN2002 12:01

208749

# 14.11.23. BIO\_L2 Listing of Immunohistochemistry Data

Listing of Persistence Results

Treatment=Treatment A

| Site<br>ID | ID/Subject | Age<br>(YEARS)/<br>Sex/<br>Race | Planned<br>Time | Date/Study<br>Day | | Interpretation | Percentage of Cells with<br>O Intensity Staining/<br>1+/ 2+/ 3+ |
|---|---|---|---|---|---|---|---|
| PPD<br>PPD | / | 65/<br>F/<br>MULTIPLE | Baseline | PPD<br>PP/ -11 | OTHER:<br>Liver | POSTIIVE | 0/<br>30/<br>10/<br>5 |
| | | | Completion/Withdrawal | <b>PPD</b> / 1 | OTHER:<br>Liver | POSTIIVE | 0/<br>30/<br>10/<br>5 |

# 208749

# 14.12. Appendix 12: Combined Preferred Terms

| Combined Term | MedDRA Preferred term | PT Code |
|---|---|---|
| | | MedDRA version 23.0 for PT codes |
| Anemia/Red blood cell count decreased | Anemia | 10002034 |
| | Red blood cell count decreased | 10038153 |
| Cytokine Release Syndrome (CRS) | Cytokine release syndrome | 10052015 |
| | Cytokine storm | 10050685 |
| Acute GVHD - Skin <sup>%</sup> | Acute graft versus host disease in skin | 10066262 |
| Acute GVHD - Gut (Liver and Intestine)% | Acute graft versus host disease in liver | 10066263 |
| | Acute graft versus host disease in intestine | 10066264 |
| Acute GVHD - Other (Lung, Bone Marrow, not specified)% | Acute graft versus host disease | 10066260 |
| Chronic GVHD - Skin <sup>%</sup> | Chronic graft versus host disease in skin | 10072159 |
| Chronic GVHD - Gut (Liver and Intestine)% | Chronic graft versus host disease in liver | 10072160 |
| | Chronic graft versus host disease in intestine | 10072158 |
| Chronic GVHD Other - (Lung, Bone Marrow, not specified) <sup>%</sup> | Chronic graft versus host disease | 10066261 |
| Unspecified GVHD - Skin <sup>%</sup> | Graft versus host disease in skin | 10064675 |
| Unspecified GVHD - Gut (Liver and Intestine) <sup>%</sup> | Graft versus host disease in liver | 10064676 |
| | Graft versus host disease in gastrointestinal tract | 10075160 |
| Unspecified GVHD - Other (Lung, Bone Marrow, not specified)% | Graft versus host disease | 10018651 |
| | Graft versus host disease in eye | 10074563 |
| | Graft versus host disease in lung | 10067742 |

208749

| Combined Term | MedDRA Preferred term | PT Code |
|---|---|---|
| | | MedDRA version 23.0 for PT codes |
| | Prophylaxis against graft versus host disease | 10053239 |
| | Transfusion associated graft versus host disease | 10070895 |
| | Engraftment syndrome | 10050684 |
| Leukopenia/White blood cell decreased | White blood cell count decreased | 10047942 |
| | Leukopenia | 10024384 |
| Lymphopenia/Lymphocyte count decreased | Lymphocyte count decreased | 10025256 |
| | CD4 lymphocytes decreased | 10007839 |
| | CD8 lymphocytes decreased | 10056283 |
| | Lymphopenia | 10025327 |
| Neutropenia/Neutrophil count decreased | Neutrophil count decreased | 10029366 |
| | Neutropenia | 10029354 |
| Rash/Rash maculo-papular | Rash maculo-papular | 10037868 |
| | Rash | 10037844 |
| | Rash erythematous | 10037855 |
| Thrombocytopenia/Platelet count decreased | Platelet count decreased | 10035528 |
| | Thrombocytopenia | 10043554 |

<sup>\*</sup> Preferred Term "RBC decreased" originally from MedDRA version 18 in Adaptimmune IB version 7 . Not in current MedDRA versions

208749

# 14.13. Appendix 13: AE Collapsing Rules

# Segments with a Common AE Preferred Term (PT) into Unique Events based on the Start and End Dates

For each unique subject, the AE records (segments) with the same AE preferred term will be collapsed into one unique AE event based on the start and end dates below.

## **Step 1 : Multiple AE Segments with Overlapped or Continuous Start/End Dates**

Multiple AE segments with a common preferred term (PT, variable=ADAE.AEDECOD) that occurred around the same time; defined as:

If a segment starts no more than one day (i.e.,  $\leq 1$  day) prior, on, or after the previous segment's end date, it is considered as an 'event'.

If the gap between the start date of a segment and the end date of previous segment is greater than one complete day (i.e., > 1 day), then consider these segments as different events.

If partial start or end dates for any AE segments, then consider these segments as separate events.

## \*\*\* NOTE: Handling of partial dates or completely missing dates

Partial dates or completely missing dates will not be imputed.

The reason for not using imputed dates is due to the small number of partial / or completely missing dates. Furthermore, using imputed dates might create additional error of up to 30 days off for the AE start or AE end dates, and can be up to 60 days off for the duration of AE.

## **Step 2: Sort Adverse Events (AE)**

For any AE event identified above:

208749

Sort the AEs segments by study ID (ADAE.STUDYID), unique subject ID (ADAE.USUBJID), AE preferred term (ADAE.AEDECOD), AE start date (ADAE.AESTDTC), and AE end date (ADAE.AEENDTC). The sorting will include all AE segments with complete or partial start / end dates.

## Step 3: Create Derived Variables in ADAE ADaM SAS Dataset

Based on the ADAE dataset sorted above under Step 2 for each unique subject, create the following derived variables in the ADAE ADaM SAS data set:

- 1) ANL01FL: Flag for the unique AE
  - a) Collapsed AE Segments

For collapsed AE segments. based on the ADAE data set sorted above under Step 2:

- derive the flag variable: ANL01FL="Y" on the first record for each collapsed AE (i.e. the earliest segment within each collapsed AE with the same ADAE.AEDECOD). In case if the AE segment of the collapsed AEs started before Lymphodepletion and ending after it, then populate the ANL01FL="Y" on very first Treatment emergent record. If there is only one record (segment) which started before lymphodepletion and ended after lymphodepletion then populate ANL01FL="Y" on that record only.
- Otherwise ANL01FL="" (Missing)
- b) AE Events Comprised of a Single Row (No Collapsing Needed)
  - derive the flag variable: ANL01FL="Y" for each single segment AE event.
- 2) EVTSEQ: Sequence number of each unique AE with the same PT

Create a sequence number, EVTSEQ, for each unique AE within the same ADAE.AEDECOD.

For each unique subject within each unique AE preferred term, this variable will be recorded as **the sequential number to identify all unique adverse events (including both single segment events (i.e., no collapsing** 

208749

# needed) and collapsed events from multiple segments) based on the sorting order chronologically addressed above under Step 2.

# a) Collapsed AE Segments

Each collapsed AE and its corresponding composed segments will have the same sequence numbers (i.e., if multiple segments/records are qualified for being collapsed into one unique AE (i.e., all those records will have same value for the derived variable EVTSEQ for that corresponding subject within the same collapsed AE).

# b) Single Segment AE Records

Each single segment AE event (i.e., un-collapsed event) will have different unique sequence number separately

# c) AE Segments with partial start or end dates

Each AE segment with partial start or end dates will have different unique sequence number starting from 99XXX, where XXX=001, 002, ...

## \* NOTE:

For those subjects who received 2 T-cell infusions, the sequential number will be based on both infusion periods combined (i.e., the assigned sequential number will be independent of T-cell infusion periods).

# Signature Page for 208749 TMF- 2069301 v 1.0

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 01-Oct-2020 17:56:16 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 01-Oct-2020 23:19:25 GMT+0000 |

Signature Page for TMF-2069301 v1.0  $\,$